CLINICAL TRIAL: NCT03299049
Title: A Phase IIIb, Randomized, Multicenter, Parallel-group, Non-inferiority, Open-label Study Evaluating the Efficacy, Safety, and Tolerability of Long-acting Cabotegravir Plus Long-acting Rilpivirine Administered Every 8 Weeks or Every 4 Weeks in HIV-1-infected Adults Who Are Virologically Suppressed
Brief Title: Efficacy, Safety and Tolerability Study of Long-acting Cabotegravir Plus Long-acting Rilpivirine (CAB LA + RPV LA) in Human-immunodeficiency Virus-1 (HIV-1) Infected Adults
Acronym: ATLAS-2M
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 207966; 2017-002946-62 (EudraCT Number)
Record Dates: First submitted 2017-09-26; First posted 2017-10-02 (Actual); Results first posted 2020-06-11 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: HIV Infections
Keywords: Long acting Cabotegravir; Safety; HIV-1; Efficacy; Tolerability; ATLAS-2M; Long acting Rilpivirine
MeSH Terms: conditions — HIV Infections | interventions — cabotegravir; Rilpivirine

STUDY DESIGN:
Intervention Model Description: Two groups of subjects will be randomized to receive CAB LA + RPV LA Q4W, or CAB LA + RPV LA Q8W regimen
Masking Description: This will be an open-label study and therefore no blinding is required
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Subjects in group 1 receiving study treatment once in 4 weeks (Experimental): Group 1 will consist of subjects randomized from current ART SOC therapy. Subjects in group 1 will be randomized to receive CAB LA plus RPV LA Q4W via intramuscular (IM) route. All subjects will receive oral therapy with CAB 30 mg + RPV 25 mg once daily prior to randomization.
  Interventions: Drug: Cabotegravir Tablets; Drug: Rilpivirine Tablets; Drug: Cabotegravir Injectable Suspension; Drug: Rilpivirine Injectable Suspension
- Subjects in group 1 receiving study treatment once in 8 weeks (Experimental): Group 1 will consist of subjects randomized from current ART SOC therapy. Subjects in group 1 will be randomized to receive CAB LA plus RPV LA Q8W via IM route. All subjects will receive oral therapy with CAB 30 mg + RPV 25 mg once daily prior to randomization.
  Interventions: Drug: Cabotegravir Tablets; Drug: Rilpivirine Tablets; Drug: Cabotegravir Injectable Suspension; Drug: Rilpivirine Injectable Suspension
- Subjects in group 2 receiving study treatment once in 4 weeks (Experimental): Group 2 will consist of subjects currently receiving CAB LA + RPV LA Q4W in ATLAS study. Subjects in Group 2 will be randomized to continue CAB LA plus RPV LA Q4W administration via IM route.
  Interventions: Drug: Cabotegravir Injectable Suspension; Drug: Rilpivirine Injectable Suspension
- Subjects in group 2 receiving study treatment once in 8 weeks (Experimental): Group 2 will consist of subjects currently receiving CAB LA + RPV LA Q4W in ATLAS study. Subjects in Group 2 will be randomized to receive CAB LA plus RPV LA Q8W via IM route.
  Interventions: Drug: Cabotegravir Injectable Suspension; Drug: Rilpivirine Injectable Suspension

INTERVENTIONS:
Drug: Cabotegravir Tablets — CAB tablets are white to almost white oval shaped film coated 30 mg tablets for oral administration. CAB tablets are to be stored up to 30 degree Celsius and protected from moisture.
  Arms: Subjects in group 1 receiving study treatment once in 4 weeks; Subjects in group 1 receiving study treatment once in 8 weeks
Drug: Rilpivirine Tablets — RPV tablets are 25 mg tablets that are off-white, round, biconvex, film-coated and debossed on one side with "TMC" and the other side with "25". RPV tablets should be stored at 25 degree Celsius (excursions permitted to 15 degree-30 degree Celsius) and protected from light.
  Arms: Subjects in group 1 receiving study treatment once in 4 weeks; Subjects in group 1 receiving study treatment once in 8 weeks
Drug: Cabotegravir Injectable Suspension — CAB LA injectable suspension is a sterile white to slightly pink suspension containing 200 mg/mL of GSK1265744 as free acid for administration by IM injection. CAB LA injectable suspension is to be stored at up to 30 degree Celsius and should not be frozen.
Drug: Rilpivirine Injectable Suspension — RPV LA injectable suspension is a sterile white suspension containing 300 mg/mL of RPV as the free base for administration by IM injection. RPV LA injectable suspension should be kept in the outer package and stored at 2-8 degree Celsius and should not be frozen. RPV LA should also be protected from light.

SUMMARY:
This Antiretroviral Therapy as Long Acting Suppression every 2 Months (ATLAS-2M) study is designed to demonstrate the non-inferior antiviral activity and safety of CAB LA + RPV LA administered every 8 weeks (Q8W) compared to CAB LA + RPV LA administered every 4 weeks (Q4W) over a 48-week treatment period in approximately 1020 adult HIV-1 infected subjects. Subjects will be divided in 2 groups; Group 1 will include subjects receiving current anti-retroviral (ART) standard of care (SOC) therapy whereas group 2 will include subjects currently receiving CAB LA + RPV LA Q4W in ATLAS study. Subjects in both groups will be randomized to receive CAB LA + RPV LA Q4W or Q8W. The study will be carried out in 3 phases including screening phase, maintenance phase and extension phase. Subjects choosing not to enter the Extension phase can complete their study participation at the Week 100 visit and enter into the 52-week Long-Term Follow-Up (LTFU) Phase as required. A sub-study in the ATLAS-2M study will evaluate the pharmacokinetics, tolerability and efficacy of CAB and RPV long acting injections following intramuscular administration in the Vastus Lateralis Muscle (thigh) in HIV-infected Adult Participants who have received at least three years of Gluteal Injections in this ATLAS-2M Study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who will be able to understand and comply with protocol requirements, instructions, and restrictions.
* Understand the long term commitment to the study and be likely to complete the study as planned
* Be considered as an appropriate candidate for participation in an investigative clinical trial with oral and intramuscularly injectable medications (e.g., no active substance use disorder, acute major organ disease, or planned long-term work assignments out of the country, etc.).
* Aged 18 years or older (or >=19 where required by local regulatory agencies), at the time of signing the informed consent.
* A female is eligible to participate if she is not pregnant (as confirmed by a negative serum human chorionic gonadotropin (hCG) test at screen and a negative urine hCG test at Randomization), not lactating, and at least one of the following conditions applies:

Non-reproductive potential defined as: pre-menopausal females with one of the following: documented tubal ligation; documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion; hysterectomy; Documented Bilateral Oophorectomy.

Postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) and estradiol levels consistent with menopause (refer to laboratory reference ranges for confirmatory levels)]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment.

Reproductive potential and agrees to follow one of the options listed in the Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) from 30 days prior to the first dose of study medication, throughout the study, for at least 30 days after discontinuation of all oral study medications, and for at least 52 weeks after discontinuation of CAB LA and RPV LA. The investigator is responsible for ensuring that participants understand how to properly use these methods of contraception.

* Capable of giving signed informed consent. Eligible subjects or their legal guardians (and next of kin when locally required), must sign a written Informed Consent Form before any protocol-specified assessments are conducted. Enrollment of subjects who are unable to provide direct informed consent is optional and will be based on local legal/regulatory requirements and site feasibility to conduct protocol procedures.
* Subjects enrolled in France must be affiliated to, or a beneficiary of, a social security category.
* Subjects receiving oral SOC treatment for HIV-1 (not participating in ATLAS Trial) must be on uninterrupted current regimen [either the initial or second anti-retroviral (ARV) regimen] for at least 6 months prior to Screening. Any prior switch, defined as a change of a single drug or multiple drugs simultaneously, must have occurred due to tolerability/safety, access to medications, or convenience/simplification, and must NOT have been done for treatment failure (HIV-1 RNA >=400 copies/mL).
* For subjects receiving oral SOC treatment for HIV-1 (not participating in ATLAS Trial) Documented evidence of at least two plasma HIV-1 RNA measurements <50 copies/mL in the 12 months prior to Screening: one within the 6 to 12-month window, and one within 6 months prior to Screening.
* For subjects receiving oral SOC treatment for HIV-1 (not participating in ATLAS Trial): Plasma HIV-1 RNA <50 copies/mL at Screening
* Subjects transitioning from 201585 (ATLAS) must have been on CAB LA 400 milligram (mg) + RPV LA 600 mg Q4W or "Current ART" regimen through at minimum Week 52 of the ATLAS study as per ATLAS protocol dosing requirements and until Day 1 of the ATLAS-2M study. Any disruptions in dosing during ATLAS must be discussed with the Medical Monitor for a final determination of eligibility.
* For Participants transitioning from 201585 (ATLAS): plasma HIV-1 RNA <50 copies/mL at Screening Sub-study inclusion criteria
* Eligible participants must have been on CAB LA + RPV LA regimen for a minimum of 152 weeks while on the ATLAS-2M study.
* Plasma HIV-1 RNA <50 c/mL at Sub-Study Screening

Exclusion Criteria:

For subjects not transitioning from 201585 (ATLAS):

* Within 6 months prior to Screening, any plasma HIV-1 RNA measurement >=50 copies/mL
* Within the 6 to 12-month window prior to Screening, any plasma HIV-1 RNA measurement >200 copies/mL, or 2 or more plasma HIV-1 RNA measurements >=50 copies/mL
* Any drug holiday during the window between initiating first HIV ART and 6 months prior to Screening, except for brief periods (less than 1 month) where all ART was stopped due to tolerability and/or safety concerns.
* Any switch to a second line regimen, defined as change of a single drug or multiple drugs simultaneously, due to virologic failure to therapy (defined as a confirmed plasma HIV 1 RNA measurement >=200 copies/mL after initial suppression to <50 copies/mL while on first line HIV therapy regimen)
* A history of use of any regimen consisting of only mono or dual HIV-1 therapy (even if only for peri-partum treatment). Subjects who are currently participating in or anticipate to be selected for any other interventional study with the exception of the 201585 (ATLAS) study.

For Subjects transitioning from 201585 (ATLAS):

* During participation in ATLAS, consecutive (2 or more sequential) plasma HIV-1 RNA measurements >=50 copies/mL
* During participation in ATLAS, any HIV-1 RNA measurement >=200 copies/mL
* More than two total measurements of plasma HIV-1 RNA >=50 c/mL during participation in the ATLAS trial will require direct approval by the ATLAS-2M Medical Monitor and Study virologist for study participation.

For all subjects:

* Women who are pregnant, breastfeeding or plan to become pregnant or breastfeed during the study.
* Any evidence of a current Center for Disease Control and Prevention (CDC) Stage 3 disease except cutaneous Kaposi's sarcoma not requiring systemic therapy and CD4+ counts <200 cells/µL are not exclusionary.
* Subjects with moderate to severe hepatic impairment.
* Any pre-existing physical or mental condition (including substance use disorder) which, in the opinion of the Investigator, may interfere with the subject's ability to comply with the dosing schedule and/or protocol evaluations or which may compromise the safety of the subject.
* Subjects determined by the Investigator to have a high risk of seizures, including participants with an unstable or poorly controlled seizure disorder. A subject with a prior history of seizure may be considered for enrollment if the Investigator believes the risk of seizure recurrence is low. All cases of prior seizure history should be discussed with the Medical Monitor prior to enrollment.
* All subjects will be screened for syphilis (rapid plasma reagin [RPR]). Subjects with untreated secondary (late latent) or tertiary syphilis infection, defined as a positive RPR and a positive treponemal test without clear documentation of treatment, are excluded. Subjects with a false positive RPR (with negative treponemal test) or serofast RPR result (persistence of a reactive nontreponemal syphilis test despite history of adequate therapy and no evidence of re-exposure) may enroll after consultation with the Medical Monitor. Participants with primary syphilis or early latent secondary syphilis (acquired within the preceding year) who have a positive RPR test and have not been treated may be treated during the screening period and if completion of antibiotic treatment occurs during the screening period, may be allowed entry after consultation with the Medical Monitor. If antibiotic treatment cannot be completed before the screening window ends, subjects may be rescreened once following completion of antibiotic therapy for primary or early latent secondary syphilis.
* Subjects who, in the investigator's judgment, pose a significant suicide risk. Subject's recent history of suicidal behavior and/or suicidal ideation should be considered when evaluating for suicide risk.
* The subject has a tattoo or other dermatological condition overlying the gluteus region which may interfere with interpretation of injection site reactions.
* Evidence of Hepatitis B virus (HBV) infection based on the results of testing at Screening for Hepatitis B surface antigen (HBsAg), Hepatitis B core antibody (anti-HBc), Hepatitis B surface antibody (anti-HBs) and HBV deoxyribonucleic acid (DNA) as follows:

Subjects positive for HBsAg are excluded; Subjects negative for anti-HBs but positive for anti-HBc (negative HBsAg status) and positive for HBV DNA are excluded. Note: Participants positive for anti-HBc (negative HBsAg status) and positive for anti-HBs (past and/or current evidence) are immune to HBV and are not excluded.

* Asymptomatic individuals with chronic hepatitis C virus (HCV) infection will not be excluded, however Investigators must carefully assess if therapy specific for HCV infection is required; participants who are anticipated to require HCV treatment within 12 months must be excluded. (HCV treatment on study may be permitted post Week 52, following consultation with the medical monitor).
* Subjects with HCV co-infection will be allowed entry into this study if: liver enzymes meet entry criteria; HCV Disease has undergone appropriate work-up, and is not advanced, and will not require treatment prior to the Week 52 visit. Additional information (where available) on participants with HCV co-infection at screening should include results from any liver biopsy, Fibroscan, ultrasound, or other fibrosis evaluation, history of cirrhosis or other decompensated liver disease, prior treatment, and timing/plan for HCV treatment; In the event that recent biopsy or imaging data is not available or inconclusive, the Fib-4 score will be used to verify eligibility: Fib-4 score >3.25 is exclusionary; Fib-4 scores 1.45 - 3.25 requires Medical Monitor consultation; Fibrosis 4 Score Formula:

(Age x AST ) / ( Platelets x ( square [ ALT ])

* Unstable liver disease (as defined by any of the following: presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice or cirrhosis), known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones or otherwise stable chronic liver disease per investigator assessment).
* History of liver cirrhosis with or without hepatitis viral co-infection.
* Ongoing or clinically relevant pancreatitis.
* Clinically significant cardiovascular disease, as defined by history/evidence of congestive heart failure, symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting (CABG) surgery or percutaneous transluminal coronary angioplasty (PTCA) or any clinically significant cardiac disease.
* Ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, non-invasive cutaneous squamous cell carcinoma, or cervical intraepithelial neoplasia; other localized malignancies require agreement between the investigator and the Study medical monitor for inclusion of the participant prior to randomization.
* Any condition which, in the opinion of the Investigator, may interfere with the absorption, distribution, metabolism or excretion of the study drugs or render the participant unable to receive study medication.
* History or presence of allergy or intolerance to the study drugs or their components or drugs of their class. In addition, if heparin is used during pharmacokinetic sampling, participants with a history of sensitivity to heparin or heparin-induced thrombocytopenia must not be enrolled.
* Current or anticipated need for chronic anti-coagulation with the exception of the use of low dose acetylsalicylic acid (<=325 mg) or hereditary coagulation and platelet disorders such as hemophilia or Von Willebrand Disease.
* Any evidence of primary resistance based on the presence of any major known Integrase inhibitor (INI) or Non-nucleoside reverse transcriptase inhibitor (NNRTI) resistance-associated mutation, except for K103N by any historical resistance test result.
* Any verified Grade 4 laboratory abnormality. A single repeat test is allowed during the Screening phase to verify a result.
* Any acute laboratory abnormality at Screening, which, in the opinion of the investigator, would preclude the subject's participation in the study of an investigational compound.
* Subjects has estimated creatine clearance <50mL/minute per 1.73 meter square (m^2) via Chronic Kidney Disease-Epidemiology Collaboration (CKD-EPI) Method
* Alanine aminotransferase (ALT) >=3 × Upper limit of normal (ULN)
* Exposure to an experimental drug (with the exception of those in the ATLAS study including CAB, CAB LA, and RPV LA) or experimental vaccine within either 30 days, 5 half-lives of the test agent, or twice the duration of the biological effect of the test agent, whichever is longer, prior to Day 1 of this study.
* Treatment with any of the following agents within 28 days of Screening: radiation therapy; cytotoxic chemotherapeutic agents; tuberculosis therapy with the exception of isoniazid (isonicotinylhydrazid, INH); anti--coagulation agents; Immunomodulators that alter immune responses such as chronic systemic corticosteroids, interleukins, or interferons. Note: Subjects using short-term (e.g. <=21 days) systemic corticosteroid treatment; topical, inhaled and intranasal corticosteroids are eligible for enrollment.
* Treatment with an HIV-1 immunotherapeutic vaccine within 90 days of Screening
* Treatment with any agent, except recognized ART as allowed above, with documented activity against HIV-1 within 28 days of study Day 1. Treatment with acyclovir/valacyclovir is permitted.
* Use of medications which are associated with Torsade de Pointes.
* Current or prior history of etravirine (ETR) use.
* Current use of tipranavir/ritonavir or fosamprenavir/ritonavir.
* Subjects receiving any prohibited medication and who are unwilling or unable to switch to an alternate medication.
* Participation in other interventional studies or non-interventional studies that require any type of assessment outside the local standard of care practices is generally not permitted, however for eligible subjects in South Africa only, co-enrolment in the AIDS Clinical Trial Group ACTG interventional study (A5392) could be exceptionally permitted after review and approval by the Medical Monitor.

Sub-study exclusion criteria

* More than 1 plasma HIV-1 RNA measurement =>50 c/mL to <200 c/mL (virologic blip) within 24 weeks prior to sub-study Screening visit.
* Any Suspected Virologic Failure (HIV-RNA>200 c/mL)
* Participants planning to require oral bridging during participation in the ATLAS-2M sub-study
* Participant has a tattoo or any dermatological condition overlying the thigh region which may interfere with interpretation of injection site reactions
* Any condition which, in the opinion of the Investigator, may interfere with the absorption, distribution, metabolism or excretion of the study drugs or render the participant unable to receive study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1049 (Actual)
Dates: Start 2017-10-27 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2029-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (94):
- United States (36):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Palm Springs, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Ft. Pierce, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, Vero Beach, Florida
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Macon, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Allentown, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Bellaire, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Longview, Texas
  - GSK Investigational Site, Annandale, Virginia
  - GSK Investigational Site, Lynchburg, Virginia
- Argentina (3):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma de Bueno
  - GSK Investigational Site, Rosario
- Australia (3):
  - GSK Investigational Site, Darlinghurst, New South Wales
  - GSK Investigational Site, Sydney, New South Wales
  - GSK Investigational Site, Prahran
- Canada (5):
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Regina, Saskatchewan
- France (5):
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Saint-Denis
  - GSK Investigational Site, Toulouse
  - GSK Investigational Site, Tourcoing
- Germany (7):
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Bonn
  - GSK Investigational Site, Essen
  - GSK Investigational Site, Frankfurt
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, Hanover
  - GSK Investigational Site, München
- Italy (2):
  - GSK Investigational Site, Brescia
  - GSK Investigational Site, Milan
- GSK Investigational Site, Guadalajara, Mexico
- Russia (11):
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Krasnodar
  - GSK Investigational Site, Lipetsk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Oryol
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, Smolensk
  - GSK Investigational Site, Toliyatti
  - GSK Investigational Site, Yekaterinburg
- South Africa (5):
  - GSK Investigational Site, Bloemfontein
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, Durban
  - GSK Investigational Site, Johannesburg
  - GSK Investigational Site, Middelburg
- South Korea (4):
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Daejeon
  - GSK Investigational Site, Pusan
  - GSK Investigational Site, Seoul
- Spain (10):
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Elche Alicante
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Vigo Pontevedra
- Sweden (2):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Background] Overton ET, Richmond G, Rizzardini G, Jaeger H, Orrell C, Nagimova F, Bredeek F, Garcia Deltoro M, Swindells S, Andrade-Villanueva JF, Wong A, Khuong-Josses MA, Van Solingen-Ristea R, van Eygen V, Crauwels H, Ford S, Talarico C, Benn P, Wang Y, Hudson KJ, Chounta V, Cutrell A, Patel P, Shaefer M, Margolis DA, Smith KY, Vanveggel S, Spreen W. Long-acting cabotegravir and rilpivirine dosed every 2 months in adults with HIV-1 infection (ATLAS-2M), 48-week results: a randomised, multicentre, open-label, phase 3b, non-inferiority study. Lancet. 2021 Dec 19;396(10267):1994-2005. doi: 10.1016/S0140-6736(20)32666-0. Epub 2020 Dec 9. PMID 33308425
- [Background] Overton ET, Richmond G, Rizzardini G, Thalme A, Girard PM, Wong A, Porteiro N, Swindells S, Reynes J, Noe S, Harrington C, Espanol CM, Acuipil C, Aksar A, Wang Y, Ford SL, Crauwels H, van Eygen V, Van Solingen-Ristea R, Latham CL, Thiagarajah S, D'Amico R, Smith KY, Vandermeulen K, Spreen WR. Long-Acting Cabotegravir and Rilpivirine Dosed Every 2 Months in Adults With Human Immunodeficiency Virus 1 Type 1 Infection: 152-Week Results From ATLAS-2M, a Randomized, Open-Label, Phase 3b, Noninferiority Study. Clin Infect Dis. 2023 May 3;76(9):1646-1654. doi: 10.1093/cid/ciad020. PMID 36660819
- [Derived] Elliot ER, Polli JW, Patel P, Garside L, Grove R, Barnett V, Roberts J, Byrapuneni S, Crauwels H, Ford SL, Van Solingen-Ristea R, Birmingham E, D'Amico R, Baugh B, van Wyk J. Efficacy, Safety, and Pharmacokinetics by Body Mass Index Category in Phase 3/3b Long-Acting Cabotegravir Plus Rilpivirine Trials. J Infect Dis. 2024 Jul 25;230(1):e34-e42. doi: 10.1093/infdis/jiad580. PMID 39052748
- [Derived] Moreno S, Rivero A, Ventayol P, Falco V, Torralba M, Schroeder M, Neches V, Vallejo-Aparicio LA, Mackenzie I, Turner M, Harrison C. Cabotegravir and Rilpivirine Long-Acting Antiretroviral Therapy Administered Every 2 Months is Cost-Effective for the Treatment of HIV-1 in Spain. Infect Dis Ther. 2023 Aug;12(8):2039-2055. doi: 10.1007/s40121-023-00840-y. Epub 2023 Jul 14. PMID 37452174
- [Derived] Chounta V, Snedecor SJ, Wu S, Van de Velde N. Indirect comparison of 48-week efficacy and safety of long-acting cabotegravir and rilpivirine maintenance every 8 weeks with daily oral standard of care antiretroviral therapy in participants with virologically suppressed HIV-1-infection. BMC Infect Dis. 2022 May 4;22(1):428. doi: 10.1186/s12879-022-07243-3. PMID 35508986
- [Derived] Jaeger H, Overton ET, Richmond G, Rizzardini G, Andrade-Villanueva JF, Mngqibisa R, Hermida AO, Thalme A, Belonosova E, Ajana F, Benn PD, Wang Y, Hudson KJ, Espanol CM, Ford SL, Crauwels H, Margolis DA, Talarico CL, Smith KY, van Eygen V, Van Solingen-Ristea R, Vanveggel S, Spreen WR. Long-acting cabotegravir and rilpivirine dosed every 2 months in adults with HIV-1 infection (ATLAS-2M), 96-week results: a randomised, multicentre, open-label, phase 3b, non-inferiority study. Lancet HIV. 2021 Nov;8(11):e679-e689. doi: 10.1016/S2352-3018(21)00185-5. Epub 2021 Oct 11. PMID 34648734
- [Derived] Swindells S, Lutz T, Van Zyl L, Porteiro N, Stoll M, Mitha E, Shon A, Benn P, Huang JO, Harrington CM, Hove K, Ford SL, Talarico CL, Chounta V, Crauwels H, Van Solingen-Ristea R, Vanveggel S, Margolis DA, Smith KY, Vandermeulen K, Spreen WR. Week 96 extension results of a Phase 3 study evaluating long-acting cabotegravir with rilpivirine for HIV-1 treatment. AIDS. 2022 Feb 1;36(2):185-194. doi: 10.1097/QAD.0000000000003025. PMID 34261093
- [Derived] Chounta V, Overton ET, Mills A, Swindells S, Benn PD, Vanveggel S, van Solingen-Ristea R, Wang Y, Hudson KJ, Shaefer MS, Margolis DA, Smith KY, Spreen WR. Patient-Reported Outcomes Through 1 Year of an HIV-1 Clinical Trial Evaluating Long-Acting Cabotegravir and Rilpivirine Administered Every 4 or 8 Weeks (ATLAS-2M). Patient. 2021 Nov;14(6):849-862. doi: 10.1007/s40271-021-00524-0. Epub 2021 May 31. PMID 34056699

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This non-inferiority study evaluated antiviral activity of cabotegravir(CAB) long acting(LA) 600 milligrams(mg) + rilpivirine(RPV) LA 900 mg administered every 8 weeks(Q8W) compared with CAB LA 400 mg+RPV LA 600 mg administered every 4 weeks(Q4W) over a 48-week period in virologically suppressed human immunodeficiency type 1 infection participants.
Pre-assignment Details: A total of 1049 eligible participants were randomized in a ratio of 1:1 to 1 of the 2 treatment arms in Maintenance Phase, of which 4 participants did not receive study treatment and 1045 participants were included in Intent to treat-Exposed Population. Results presented are based on Week 48 primary analysis.
Groups:
- CAB LA + RPV LA Q8W: Eligible participants transitioning from antiretroviral (ART) standard of care (SOC) therapy arm and CAB LA + RPV LA Q4W arm in the ATLAS (NCT02951052) study and randomized to receive CAB LA+RPV LA Q8W in the current study were administered oral therapy with CAB 30 mg + RPV 25 mg once daily at Day 1 for 4 weeks. Participants then received intramuscular (IM) injections of CAB LA 600 mg and RPV LA 900 mg at Week 4b and Week 8 followed by injections Q8W thereafter. Participants transitioned from the CAB LA+RPV LA Q4W arm of ATLAS study received CAB LA 600 mg+RPV LA 900 mg intramuscular injections on Day 1, Week 8 and Q8W thereafter.
- CAB LA + RPV LA Q4W: Eligible participants transitioning from ART SOC arm and CAB LA + RPV LA Q4W arm in the ATLAS (NCT02951052) study and randomized to receive CAB LA+RPV LA Q4W in the current study were administered oral therapy with CAB 30 mg + RPV 25 mg once daily at Day 1 for 4 weeks. Participants then received a loading dose of CAB LA 600 mg and RPV LA 900 mg IM injections at Week 4b followed maintenance injections of CAB LA 400 mg +RPV LA 600 mg Q4W thereafter. Participants transitioned from the Q4W arm of ATLAS study continued to receive CAB LA 400 mg+RPV LA 600 mg intramuscular injections administered Q4W from Day 1.
Period: Overall Study
Arm/Group | CAB LA + RPV LA Q8W | CAB LA + RPV LA Q4W
Started | 522 | 523
Completed | 0 | 0
Not Completed | 522 | 523
Not completed — On-going | 486 | 481
Not completed — Withdrawal by Subject | 6 | 21
Not completed — Physician Decision | 5 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Pregnancy | 1 | 3
Not completed — Protocol Violation | 1 | 1
Not completed — Lack of Efficacy | 9 | 3
Not completed — Adverse Event | 12 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CAB LA + RPV LA Q8W | CAB LA + RPV LA Q4W | Total
Number analyzed (Participants) | 522 | 523 | 1045
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.7 (11.16) | 42.3 (10.58) | 42.5 (10.87)
Sex/Gender, Customized [Number; unit: Participants]
  Sex at birth=Female | 137 | 143 | 280
  Sex at birth=Male | 385 | 380 | 765
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Reported gender=Female | 142 | 146 | 288
  Reported gender=Male | 380 | 377 | 757
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian (AI) or Alaska Native (AN) | 17 | 11 | 28
  Asian-Central/South Asian Heritage (H) | 1 | 1 | 2
  Asian-East Asian H | 20 | 12 | 32
  Asian-Japanese H | 0 | 2 | 2
  Asian-South East Asian (SEA) H | 8 | 7 | 15
  Black or African American (AA) | 101 | 90 | 191
  Native Hawaiian (NH) or other Pacific Islander | 3 | 1 | 4
  White-Arabic/North African H | 2 | 4 | 6
  White-White/Caucasian/European (EU) H | 368 | 388 | 756
  White-Mixed White Race | 0 | 1 | 1
  Multiple-AI/AN and Black/AA/White/Caucasian/EU H | 1 | 1 | 2
  Multiple-AI/AN and NH/Other Pacific Islander | 1 | 0 | 1
  Multiple-SEA H and White/Caucasian/ EU H | 0 | 1 | 1
  Multiple-Black/AA and White-Arabic/North African H | 0 | 1 | 1
  Multiple-Black/AA and White/Caucasian/EU H | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Plasma Human Immunodeficiency Virus-ribonucleic Acid (HIV-RNA) >=50 Copies Per Milliliter (c/mL) as Per Food and Drug Administration (FDA) Snapshot Algorithm at Week 48
Description: Percentage of participants with HIV-1 RNA >=50 c/mL as per FDA snapshot algorithm at Week 48 was assessed to demonstrate the non-inferior antiviral activity of CAB LA+RPV LA Q8W compared to CAB LA + RPV LA Q4W regimen over 48 weeks in HIV-1 infected ART experienced participants. The HIV-1 RNA >=50 c/mL per Snapshot algorithm was determined by the last on-treatment HIV-1 RNA measurement within the Week 48 analysis visit window. Intent-to-treat-Exposed (ITT-E) Population comprised of all randomized participants who received at least one dose of study treatment. Participants were assessed according to their randomized treatment, regardless of the treatment they received.
Time Frame: Week 48
Population: ITT-E Population.
Measure: Number; unit: Percentage of participants
Arm/Group | CAB LA + RPV LA Q8W | CAB LA + RPV LA Q4W
Number analyzed (Participants) | 522 | 523
Percentage of participants | 1.7 | 1.0
Statistical Analysis 1: Comparison: CAB LA + RPV LA Q8W vs CAB LA + RPV LA Q4W; Test type: Non-Inferiority — Non-inferiority was concluded if the upper bound of the two-sided 95% confidence interval (CI) for the Cochran-Mantel Haenzel (CMH) adjusted treatment difference (Q8W minus Q4W) is less than 4%; Adjusted difference = 0.8, 95% CI 2-sided [-0.6 to 2.2] — Adjusted CMH estimate of the difference in the percentage of participants with Plasma HIV-1 >=50 c/mL between each treatment group (Q8W - Q4W) and corresponding 95% CI is presented

2. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA <50 c/mL Using FDA Snapshot Algorithm at Week 48
Description: Percentage of participants with plasma HIV-1 RNA <50 c/mL at Week 48 using FDA Snapshot algorithm was assessed to demonstrate antiviral activity of CAB LA+RPV LA Q8W compared to CAB LA+ RPV LA Q4W. The HIV-1 RNA <50 c/mL per Snapshot algorithm was determined by last on-treatment HIV-1 RNA measurement within the analysis visit window. The 95% CIs were derived using normal approximation (Wald CI)
Time Frame: Week 48
Population: ITT-E Population.
Measure: Number; unit: Percentage of participants
Arm/Group | CAB LA + RPV LA Q8W | CAB LA + RPV LA Q4W
Number analyzed (Participants) | 522 | 523
Percentage of participants | 94 | 93
Statistical Analysis 1: Comparison: CAB LA + RPV LA Q8W vs CAB LA + RPV LA Q4W; Test type: Non-Inferiority — Non-inferiority was concluded if the upper bound of the two-sided 95% CI for the CMH adjusted treatment difference (Q8W minus Q4W) is greater than -10%; Adjusted difference = 0.8, 95% CI 2-sided [-2.1 to 3.7] — Adjusted CMH estimate of the difference in the percentage of participants with Plasma HIV-1 <50 c/mL between each treatment group (Q8W-Q4W) and corresponding 95% CI is presented

3. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA <50 c/mL Using FDA Snapshot Algorithm at Week 24
Description: as for outcome 2
Time Frame: Week 24
Population: ITT-E Population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CAB LA + RPV LA Q8W | CAB LA + RPV LA Q4W
Number analyzed (Participants) | 522 | 523
Percentage of participants | 95 [93 to 97] | 95 [94 to 97]

4. Secondary Outcome: Percentage of Participants With Protocol Defined Confirmed Virologic Failure (CVF) Through Weeks 24 and 48
Description: CVF was defined as rebound as indicated by two consecutive plasma HIV-1-RNA levels >=200 c/mL after prior suppression to <200 c/mL. Cumulative percentage of participants with protocol defined CVF up to Weeks 24 and 48 has been presented.
Time Frame: Weeks 24 and 48
Population: ITT-E Population.
Measure: Number; unit: Percentage of participants
Arm/Group | CAB LA + RPV LA Q8W | CAB LA + RPV LA Q4W
Number analyzed (Participants) | 522 | 523
Percentage of participants
  Week 24 | 1.3 | 0.2
  Week 48 | 1.5 | 0.4

5. Secondary Outcome: Percentage of Participants With HIV-RNA >=50 c/mL as Per FDA Snapshot Algorithm at Week 24
Description: Percentage of participants with plasma HIV-1 RNA >=50 c/mL at Week 24 using FDA Snapshot algorithm was assessed to demonstrate antiviral activity of CAB LA+RPV LA Q8W compared to CAB LA+ RPV LA Q4W. The HIV-1 RNA >=50 c/mL per Snapshot algorithm was determined by the last on-treatment HIV-1 RNA measurement within the analysis visit window. The 95% CIs were derived using normal approximation (Wald CI).
Time Frame: Weeks 24
Population: ITT-E Population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CAB LA + RPV LA Q8W | CAB LA + RPV LA Q4W
Number analyzed (Participants) | 522 | 523
Percentage of participants | 2.1 [0.9 to 3.3] | 1.5 [0.5 to 2.6]

6. Secondary Outcome: Absolute Values for HIV-1 RNA at Week 48
Description: Plasma samples were collected for quantitative analysis of HIV-1 RNA. Logarithm to base 10 (log10) values for plasma HIV-1 RNA has been presented.
Time Frame: Weeks 48
Population: ITT-E Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Log 10 c/mL
Arm/Group | CAB LA + RPV LA Q8W | CAB LA + RPV LA Q4W
Number analyzed (Participants) | 493 | 487
Log 10 c/mL | 1.599 (0.0870) | 1.593 (0.0302)

7. Secondary Outcome: Change From Baseline Values for HIV-1 RNA at Week 48
Description: Plasma samples were collected for quantitative analysis of HIV-1 RNA. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is defined as post-dose visit value minus Baseline value. Logarithm to base 10 values for plasma HIV-1 RNA has been presented.
Time Frame: Baseline (Day 1) and Week 48
Population: ITT-E Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Log 10 c/mL
Arm/Group | CAB LA + RPV LA Q8W | CAB LA + RPV LA Q4W
Number analyzed (Participants) | 493 | 487
Log 10 c/mL | 0.007 (0.0888) | -0.015 (0.1673)

8. Secondary Outcome: Absolute Values for Cluster of Differentiation 4 Plus (CD4+) at Week 48
Description: Blood samples were collected and CD4+ cell count assessment by flow cytometry was carried out to evaluate the immunologic activity of CAB LA+RPV LA Q8W compared to CAB LA+RPV LA Q8W.
Time Frame: Week 48
Population: ITT-E Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Cells per cubic millimeter
Arm/Group | CAB LA + RPV LA Q8W | CAB LA + RPV LA Q4W
Number analyzed (Participants) | 493 | 486
Cells per cubic millimeter | 685.9 (261.70) | 700.0 (278.18)

9. Secondary Outcome: Change From Baseline Values for CD4+ at Week 48
Description: Blood samples were collected and CD4+ cell count assessment by flow cytometry was carried out to evaluate the immunologic activity of CAB LA+RPV LA Q8W compared to CAB LA+RPV LA Q4W. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and Week 48
Population: ITT-E Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Cells per cubic millimeter
Arm/Group | CAB LA + RPV LA Q8W | CAB LA + RPV LA Q4W
Number analyzed (Participants) | 493 | 486
Cells per cubic millimeter | 5.3 (168.62) | -24.6 (199.02)

10. Secondary Outcome: Number of Participants With Non-serious Adverse Events (Non-SAEs >=5% Incidence) and Serious Adverse Events (SAEs)-Maintenance Phase
Description: An adverse event is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. A SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect, associated with liver injury and impaired liver function or any other situations as per medical or scientific judgement. Safety Population comprised of all randomized participants who received at least one dose of study treatment. Participants were assessed according to actual treatment received.
Time Frame: Up to Week 48
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA + RPV LA Q8W | CAB LA + RPV LA Q4W
Number analyzed (Participants) | 522 | 523
Participants
  Any non-SAE (>=5%) | 429 | 427
  Any SAE | 27 | 19

11. Secondary Outcome: Number of Participants With Severity of Adverse Events-Maintenance Phase
Description: Severity of adverse events were defined as per The Division of Acquired Immunodeficiency Syndrome (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS adverse events Grading Table). Severity grades for adverse events were as Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), Grade 4 (Potentially life-threatening) and Grade 5 (all deaths related to an AE).
Time Frame: Up to Week 48
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA + RPV LA Q8W | CAB LA + RPV LA Q4W
Number analyzed (Participants) | 522 | 523
Participants
  Grade 1 | 201 | 195
  Grade 2 | 231 | 238
  Grade 3 | 38 | 43
  Grade 4 | 2 | 6
  Grade 5 | 1 | 0

12. Secondary Outcome: Number of Participants With Maximum Post-Baseline Chemistry Toxicities-Maintenance Phase
Description: Clinical chemistry toxicities were graded as per the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table)Blood samples were collected for the analysis of following clinical chemistry parameters: alanine aminotransferase (ALT), albumin, alkaline phosphate (ALP), aspartate aminotranferase (AST), bilirubin, carbon dioxide (CO2), cholesterol, creatinine kinase, creatinine, glomerular filtration rate (GFR) from creatinine adjusted for bovine serum albumin (BSA), glucose, hyperglycemia, hyperkalemia, hypernatremia, hypoglycemia, hypokalemia, hyponatremia, low density lipoprotein (LDL) calculation, lipase, phosphate, potassium, sodium and triglycerides. Severity grades were: Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe) and Grade 4 (Potentially life-threatening).
Time Frame: Up to Week 48
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA + RPV LA Q8W | CAB LA + RPV LA Q4W
Number analyzed (Participants) | 522 | 523
Participants
  ALT, Grade 1 | 45 | 49
  ALT, Grade 2 | 10 | 13
  ALT, Grade 3 | 1 | 3
  ALT, Grade 4 | 1 | 2
  Albumin, Grade 1 | 1 | 0
  Albumin, Grade 2 | 1 | 1
  Albumin, Grade 3 | 0 | 0
  Albumin, Grade 4 | 0 | 0
  ALP, Grade 1 | 1 | 5
  ALP, Grade 2 | 0 | 0
  ALP, Grade 3 | 0 | 0
  ALP, Grade 4 | 0 | 0
  AST, Grade 1 | 32 | 44
  AST, Grade 2 | 10 | 13
  AST, Grade 3 | 2 | 4
  AST, Grade 4 | 1 | 2
  Bilirubin, Grade 1 | 27 | 25
  Bilirubin, Grade 2 | 7 | 5
  Bilirubin, Grade 3 | 1 | 1
  Bilirubin, Grade 4 | 1 | 1
  CO2, Grade 1 | 98 | 111
  CO2, Grade 2 | 2 | 1
  CO2, Grade 3 | 0 | 0
  CO2, Grade 4 | 0 | 0
  Cholesterol, Grade 1 | 50 | 52
  Cholesterol, Grade 2 | 31 | 30
  Cholesterol, Grade 3 | 2 | 3
  Cholesterol, Grade 4 | 0 | 0
  Creatinine Kinase, Grade 1 | 41 | 32
  Creatinine Kinase, Grade 2 | 22 | 19
  Creatinine Kinase, Grade 3 | 7 | 9
  Creatinine Kinase, Grade 4 | 9 | 14
  Creatinine, Grade 1 | 5 | 9
  Creatinine, Grade 2 | 2 | 1
  Creatinine, Grade 3 | 0 | 0
  Creatinine, Grade 4 | 0 | 0
  GFR from creatinine adjusted for BSA, Grade 1 | 0 | 0
  GFR from creatinine adjusted for BSA, Grade 2 | 110 | 134
  GFR from creatinine adjusted for BSA, Grade 3 | 15 | 19
  GFR from creatinine adjusted for BSA, Grade 4 | 0 | 1
  Glucose, Grade 1 | 84 | 87
  Glucose, Grade 2 | 34 | 43
  Glucose, Grade 3 | 3 | 5
  Glucose, Grade 4 | 1 | 1
  Hyperglycemia, Grade 1 | 80 | 77
  Hyperglycemia, Grade 2 | 32 | 38
  Hyperglycemia, Grade 3 | 2 | 5
  Hyperglycemia, Grade 4 | 0 | 0
  Hyperkalemia, Grade 1 | 8 | 2
  Hyperkalemia, Grade 2 | 0 | 1
  Hyperkalemia, Grade 3 | 0 | 0
  Hyperkalemia, Grade 4 | 0 | 1
  Hypernatremia, Grade 1 | 6 | 2
  Hypernatremia, Grade 2 | 0 | 0
  Hypernatremia, Grade 3 | 0 | 0
  Hypernatremia, Grade 4 | 0 | 0
  Hypoglycemia, Grade 1 | 11 | 13
  Hypoglycemia, Grade 2 | 2 | 5
  Hypoglycemia, Grade 3 | 1 | 0
  Hypoglycemia, Grade 4 | 1 | 1
  Hypokalemia, Grade 1 | 10 | 8
  Hypokalemia, Grade 2 | 0 | 0
  Hypokalemia, Grade 3 | 0 | 0
  Hypokalemia, Grade 4 | 0 | 0
  Hyponatremia, Grade 1 | 23 | 26
  Hyponatremia, Grade 2 | 0 | 1
  Hyponatremia, Grade 3 | 0 | 0
  Hyponatremia, Grade 4 | 0 | 0
  LDL Cholesterol calculation, Grade 1 | 40 | 41
  LDL Cholesterol calculation, Grade 2 | 20 | 26
  LDL Cholesterol calculation, Grade 3 | 9 | 4
  LDL Cholesterol calculation, Grade 4 | 0 | 0
  Lipase, Grade 1 | 40 | 44
  Lipase, Grade 2 | 31 | 44
  Lipase, Grade 3 | 13 | 4
  Lipase, Grade 4 | 3 | 6
  Phosphate, Grade 1 | 75 | 72
  Phosphate, Grade 2 | 20 | 1
  Phosphate, Grade 3 | 0 | 2
  Phosphate, Grade 4 | 0 | 0
  Potassium, Grade 1 | 18 | 10
  Potassium, Grade 2 | 0 | 1
  Potassium, Grade 3 | 0 | 0
  Potassium, Grade 4 | 0 | 1
  Sodium, Grade 1 | 29 | 28
  Sodium, Grade 2 | 0 | 1
  Sodium, Grade 3 | 0 | 0
  Sodium, Grade 4 | 0 | 0
  Triglycerides, Grade 1 | 51 | 42
  Triglycerides, Grade 2 | 11 | 3
  Triglycerides, Grade 3 | 4 | 2
  Triglycerides, Grade 4 | 0 | 2

13. Secondary Outcome: Number of Participants With Maximum Post-Baseline Hematology Toxicities-Maintenance Phase
Description: The hematology toxicities were graded as per the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table). Blood samples were collected for the analysis of following hematology parameters: hemoglobin, leukocytes, neutrophils and platelets. Severity grades were as Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe) and Grade 4 (Potentially life-threatening).
Time Frame: Up to Week 48
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA + RPV LA Q8W | CAB LA + RPV LA Q4W
Number analyzed (Participants) | 522 | 523
Participants
  Hemoglobin, Grade 1 | 9 | 4
  Hemoglobin, Grade 2 | 1 | 3
  Hemoglobin, Grade 3 | 2 | 4
  Hemoglobin, Grade 4 | 0 | 0
  Leukocytes, Grade 1 | 12 | 5
  Leukocytes, Grade 2 | 0 | 0
  Leukocytes, Grade 3 | 1 | 0
  Leukocytes, Grade 4 | 0 | 0
  Neutrophils, Grade 1 | 7 | 6
  Neutrophils, Grade 2 | 8 | 5
  Neutrophils, Grade 3 | 1 | 2
  Neutrophils, Grade 4 | 2 | 1
  Platelets, Grade 1 | 8 | 8
  Platelets, Grade 2 | 1 | 1
  Platelets, Grade 3 | 1 | 1
  Platelets, Grade 4 | 0 | 0

14. Secondary Outcome: Percentage of Participants Who Discontinued Treatment Due to Adverse Events-Maintenance Phase
Description: An adverse event is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. Percentage of participants with adverse events leading to withdrawal has been presented.
Time Frame: Up to Week 48
Population: Safety Population.
Measure: Number; unit: Percentage of participants
Arm/Group | CAB LA + RPV LA Q8W | CAB LA + RPV LA Q4W
Number analyzed (Participants) | 522 | 523
Percentage of participants | 2 | 2

15. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: ALT, ALP, AST and Creatinine Kinase Over Time
Description: Blood samples were collected for the analysis of clinical chemical parameters including ALT, ALP, AST and creatinine kinase. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and Weeks 4, 8, 16, 24, 32, 40 and 48
Population: Safety Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | CAB LA + RPV LA Q8W | CAB LA + RPV LA Q4W
Number analyzed (Participants) | 522 | 523
International units per liter
  ALT, Week 4, n=326, 520: number analyzed (Participants) | 326 | 520
  ALT, Week 4, n=326, 520 | -1.3 (11.11) | 0.1 (14.01)
  ALT, Week 8, n=510, 515: number analyzed (Participants) | 510 | 515
  ALT, Week 8, n=510, 515 | 0.8 (21.28) | 0.3 (15.65)
  ALT, Week 16, n=515, 513: number analyzed (Participants) | 515 | 513
  ALT, Week 16, n=515, 513 | 1.5 (47.60) | -0.7 (12.29)
  ALT, Week 24, n=505, 503: number analyzed (Participants) | 505 | 503
  ALT, Week 24, n=505, 503 | 1.9 (63.03) | -0.3 (13.39)
  ALT, Week 32, n=499, 498: number analyzed (Participants) | 499 | 498
  ALT, Week 32, n=499, 498 | -0.4 (12.60) | 2.4 (33.72)
  ALT, Week 40, n=495, 490: number analyzed (Participants) | 495 | 490
  ALT, Week 40, n=495, 490 | 0.4 (13.50) | 6.6 (112.13)
  ALT, Week 48, n=493, 486: number analyzed (Participants) | 493 | 486
  ALT, Week 48, n=493, 486 | 1.1 (16.39) | 1.6 (18.61)
  ALP, Week 4, n=326, 520: number analyzed (Participants) | 326 | 520
  ALP, Week 4, n=326, 520 | -5.5 (12.09) | -2.1 (10.25)
  ALP, Week 8, n=510, 515: number analyzed (Participants) | 510 | 515
  ALP, Week 8, n=510, 515 | -4.1 (13.07) | -3.3 (11.31)
  ALP, Week 16, n=515, 513: number analyzed (Participants) | 515 | 513
  ALP, Week 16, n=515, 513 | -4.8 (14.65) | -4.2 (13.07)
  ALP, Week 24, n=505, 503: number analyzed (Participants) | 505 | 503
  ALP, Week 24, n=505, 503 | -5.2 (16.04) | -4.0 (13.42)
  ALP, Week 32, n=499, 498: number analyzed (Participants) | 499 | 498
  ALP, Week 32, n=499, 498 | -5.7 (17.14) | -4.1 (14.95)
  ALP, Week 40, n=495, 490: number analyzed (Participants) | 495 | 490
  ALP, Week 40, n=495, 490 | -5.9 (17.61) | -3.9 (16.09)
  ALP, Week 48, n=493, 486: number analyzed (Participants) | 493 | 486
  ALP, Week 48, n=493, 486 | -6.6 (17.18) | -4.5 (15.02)
  AST, Week 4, n=326, 520: number analyzed (Participants) | 326 | 520
  AST, Week 4, n=326, 520 | -0.6 (13.25) | -0.3 (18.47)
  AST, Week 8, n=510, 515: number analyzed (Participants) | 510 | 515
  AST, Week 8, n=510, 515 | 0.6 (11.71) | 0.0 (14.46)
  AST, Week 16, n=515, 513: number analyzed (Participants) | 515 | 513
  AST, Week 16, n=515, 513 | 1.2 (24.79) | -0.3 (16.58)
  AST, Week 24, n=505, 503: number analyzed (Participants) | 505 | 503
  AST, Week 24, n=505, 503 | 1.6 (53.81) | -0.2 (21.65)
  AST, Week 32, n=499, 498: number analyzed (Participants) | 499 | 498
  AST, Week 32, n=499, 498 | -1.6 (8.84) | 0.8 (34.81)
  AST, Week 40, n=495, 490: number analyzed (Participants) | 495 | 490
  AST, Week 40, n=495, 490 | -1.0 (10.14) | 2.5 (66.54)
  AST, Week 48, n=493, 486: number analyzed (Participants) | 493 | 486
  AST, Week 48, n=493, 486 | -0.2 (12.48) | -0.7 (16.12)
  Creatinine kinase, Week 4, n=326, 520: number analyzed (Participants) | 326 | 520
  Creatinine kinase, Week 4, n=326, 520 | 30.2 (689.41) | -29.3 (717.51)
  Creatinine kinase, Week 8, n=510, 515: number analyzed (Participants) | 510 | 515
  Creatinine kinase, Week 8, n=510, 515 | 24.1 (479.84) | -23.7 (682.90)
  Creatinine kinase, Week 16, n=515, 513: number analyzed (Participants) | 515 | 513
  Creatinine kinase, Week 16, n=515, 513 | 30.6 (692.65) | -4.7 (856.65)
  Creatinine kinase, Week 24, n=505, 503: number analyzed (Participants) | 505 | 503
  Creatinine kinase, Week 24, n=505, 503 | -13.6 (265.16) | 31.1 (1198.22)
  Creatinine kinase, Week 32, n=499, 498: number analyzed (Participants) | 499 | 498
  Creatinine kinase, Week 32, n=499, 498 | -23.3 (314.46) | -5.8 (787.02)
  Creatinine kinase, Week 40, n=495, 490: number analyzed (Participants) | 495 | 490
  Creatinine kinase, Week 40, n=495, 490 | -12.5 (336.08) | 34.2 (1288.66)
  Creatinine kinase, Week 48, n=493, 486: number analyzed (Participants) | 493 | 486
  Creatinine kinase, Week 48, n=493, 486 | 17.9 (411.70) | -2.9 (810.46)

16. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter: Albumin Over Time
Description: Blood samples were collected for the analysis of clinical chemistry parameter: albumin. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and Weeks 4, 8, 16, 24, 32, 40 and 48
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | CAB LA + RPV LA Q8W | CAB LA + RPV LA Q4W
Number analyzed (Participants) | 522 | 523
Grams per liter
  Week 4, n=326, 520: number analyzed (Participants) | 326 | 520
  Week 4, n=326, 520 | -0.5 (2.32) | -0.2 (2.45)
  Week 8, n=510, 515: number analyzed (Participants) | 510 | 515
  Week 8, n=510, 515 | -0.3 (2.48) | -0.1 (2.48)
  Week 16, n=515, 513: number analyzed (Participants) | 515 | 513
  Week 16, n=515, 513 | -0.3 (2.56) | -0.4 (2.51)
  Week 24, n=505, 503: number analyzed (Participants) | 505 | 503
  Week 24, n=505, 503 | -0.0 (2.49) | -0.2 (2.59)
  Week 32, n=499, 498: number analyzed (Participants) | 499 | 498
  Week 32, n=499, 498 | -0.2 (2.63) | -0.3 (2.68)
  Week 40, n=495, 490: number analyzed (Participants) | 495 | 490
  Week 40, n=495, 490 | 0.1 (2.68) | -0.3 (2.54)
  Week 48, n=493, 486: number analyzed (Participants) | 493 | 486
  Week 48, n=493, 486 | -0.2 (2.59) | -0.2 (2.60)

17. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Bilirubin and Creatinine Over Time
Description: Blood samples were collected for the analysis of clinical chemistry parameters: bilirubin and creatinine. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and Weeks 4, 8, 16, 24, 32, 40 and 48
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | CAB LA + RPV LA Q8W | CAB LA + RPV LA Q4W
Number analyzed (Participants) | 522 | 523
Micromoles per liter
  Bilirubin, Week 4, n=326, 520: number analyzed (Participants) | 326 | 520
  Bilirubin, Week 4, n=326, 520 | 0.4 (6.44) | 0.1 (5.70)
  Bilirubin, Week 8, n=510, 515: number analyzed (Participants) | 510 | 515
  Bilirubin, Week 8, n=510, 515 | 0.4 (5.68) | 0.1 (5.39)
  Bilirubin, Week 16, n=515, 513: number analyzed (Participants) | 515 | 513
  Bilirubin, Week 16, n=515, 513 | 0.5 (5.78) | 0.2 (5.69)
  Bilirubin, Week 24, n=505, 503: number analyzed (Participants) | 505 | 503
  Bilirubin, Week 24, n=505, 503 | 0.8 (9.42) | 0.5 (5.23)
  Bilirubin, Week 32, n=499, 498: number analyzed (Participants) | 499 | 498
  Bilirubin, Week 32, n=499, 498 | 0.5 (5.54) | 0.4 (5.46)
  Bilirubin, Week 40, n=495, 490: number analyzed (Participants) | 495 | 490
  Bilirubin, Week 40, n=495, 490 | 0.7 (6.00) | 0.4 (5.77)
  Bilirubin, Week 48, n=493, 486: number analyzed (Participants) | 493 | 486
  Bilirubin, Week 48, n=493, 486 | 0.4 (5.77) | 0.7 (4.93)
  Creatinine, Week 4, n=326, 521: number analyzed (Participants) | 326 | 521
  Creatinine, Week 4, n=326, 521 | 0.89 (8.768) | -0.36 (7.215)
  Creatinine, Week 8, n=510, 515: number analyzed (Participants) | 510 | 515
  Creatinine, Week 8, n=510, 515 | -0.94 (8.638) | -0.39 (8.191)
  Creatinine, Week 16, n=515, 513: number analyzed (Participants) | 515 | 513
  Creatinine, Week 16, n=515, 513 | -0.24 (8.973) | -0.03 (8.516)
  Creatinine, Week 24, n=505, 503: number analyzed (Participants) | 505 | 503
  Creatinine, Week 24, n=505, 503 | 0.22 (9.085) | 0.94 (9.591)
  Creatinine, Week 32, n=499, 498: number analyzed (Participants) | 499 | 498
  Creatinine, Week 32, n=499, 498 | 1.01 (9.490) | 2.09 (9.313)
  Creatinine, Week 40, n=495, 490: number analyzed (Participants) | 495 | 490
  Creatinine, Week 40, n=495, 490 | 1.02 (9.604) | 2.05 (9.414)
  Creatinine, Week 48, n=493, 486: number analyzed (Participants) | 493 | 486
  Creatinine, Week 48, n=493, 486 | 1.30 (9.813) | 2.30 (8.678)

18. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: CO2, Chloride, Phosphate, Potassium, Sodium and Urea Over Time
Description: Blood samples were collected for the analysis of clinical chemistry parameters: CO2, chloride, phosphate, potassium, sodium and urea. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and Weeks 4, 8, 16, 24, 32, 40 and 48
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | CAB LA + RPV LA Q8W | CAB LA + RPV LA Q4W
Number analyzed (Participants) | 522 | 523
Millimoles per liter
  CO2, Week 4, n=326, 520: number analyzed (Participants) | 326 | 520
  CO2, Week 4, n=326, 520 | -0.5 (2.29) | -0.7 (2.32)
  CO2, Week 8, n=510, 515: number analyzed (Participants) | 510 | 515
  CO2, Week 8, n=510, 515 | -0.8 (2.12) | -0.8 (2.23)
  CO2, Week 16, n=515, 513: number analyzed (Participants) | 515 | 513
  CO2, Week 16, n=515, 513 | -1.0 (2.31) | -0.9 (2.33)
  CO2, Week 24, n=505, 503: number analyzed (Participants) | 505 | 503
  CO2, Week 24, n=505, 503 | -0.7 (2.38) | -0.7 (2.28)
  CO2, Week 32, n=499, 498: number analyzed (Participants) | 499 | 498
  CO2, Week 32, n=499, 498 | -0.9 (2.31) | -0.8 (2.43)
  CO2, Week 40, n=495, 490: number analyzed (Participants) | 495 | 490
  CO2, Week 40, n=495, 490 | -0.6 (2.33) | -0.7 (2.44)
  CO2, Week 48, n=493, 485: number analyzed (Participants) | 493 | 485
  CO2, Week 48, n=493, 485 | -0.4 (2.32) | -0.4 (2.41)
  Chloride, Week 4, n=326, 520: number analyzed (Participants) | 326 | 520
  Chloride, Week 4, n=326, 520 | 0.6 (2.19) | 0.2 (2.35)
  Chloride, Week 8, n=510, 515: number analyzed (Participants) | 510 | 515
  Chloride, Week 8, n=510, 515 | 0.3 (2.24) | 0.2 (2.34)
  Chloride, Week 16, n=515, 513: number analyzed (Participants) | 515 | 513
  Chloride, Week 16, n=515, 513 | 0.4 (2.30) | 0.2 (2.40)
  Chloride, Week 24, n=505, 503: number analyzed (Participants) | 505 | 503
  Chloride, Week 24, n=505, 503 | 0.1 (2.36) | -0.1 (2.59)
  Chloride, Week 32, n=499, 498: number analyzed (Participants) | 499 | 498
  Chloride, Week 32, n=499, 498 | 0.2 (2.34) | 0.1 (2.64)
  Chloride, Week 40, n=495, 490: number analyzed (Participants) | 495 | 490
  Chloride, Week 40, n=495, 490 | -0.1 (2.46) | 0.0 (2.36)
  Chloride, Week 48, n=493, 486: number analyzed (Participants) | 493 | 486
  Chloride, Week 48, n=493, 486 | -0.0 (2.25) | -0.1 (2.46)
  Phosphate, Week 4, n=326, 520: number analyzed (Participants) | 326 | 520
  Phosphate, Week 4, n=326, 520 | 0.054 (0.182) | 0.018 (0.167)
  Phosphate, Week 8, n=510, 515: number analyzed (Participants) | 510 | 515
  Phosphate, Week 8, n=510, 515 | 0.025 (0.177) | 0.029 (0.160)
  Phosphate, Week 16, n=515, 513: number analyzed (Participants) | 515 | 513
  Phosphate, Week 16, n=515, 513 | 0.017 (0.181) | 0.007 (0.172)
  Phosphate, Week 24, n=505, 502: number analyzed (Participants) | 505 | 502
  Phosphate, Week 24, n=505, 502 | 0.016 (0.170) | -0.004 (0.168)
  Phosphate, Week 32, n=499, 498: number analyzed (Participants) | 499 | 498
  Phosphate, Week 32, n=499, 498 | -0.001 (0.183) | 0.001 (0.172)
  Phosphate, Week 40, n=495, 490: number analyzed (Participants) | 495 | 490
  Phosphate, Week 40, n=495, 490 | 0.014 (0.180) | 0.001 (0.170)
  Phosphate, Week 48, n=493, 486: number analyzed (Participants) | 493 | 486
  Phosphate, Week 48, n=493, 486 | 0.007 (0.169) | 0.010 (0.157)
  Potassium, Week 4, n=326, 520: number analyzed (Participants) | 326 | 520
  Potassium, Week 4, n=326, 520 | 0.03 (0.337) | 0.03 (0.303)
  Potassium, Week 8, n=510, 515: number analyzed (Participants) | 510 | 515
  Potassium, Week 8, n=510, 515 | 0.04 (0.317) | 0.04 (0.331)
  Potassium, Week 16, n=515, 513: number analyzed (Participants) | 515 | 513
  Potassium, Week 16, n=515, 513 | 0.03 (0.328) | 0.03 (0.341)
  Potassium, Week 24, n=505, 503: number analyzed (Participants) | 505 | 503
  Potassium, Week 24, n=505, 503 | 0.04 (0.338) | 0.03 (0.321)
  Potassium, Week 32, n=499, 498: number analyzed (Participants) | 499 | 498
  Potassium, Week 32, n=499, 498 | 0.04 (0.364) | 0.00 (0.340)
  Potassium, Week 40, n=495, 490: number analyzed (Participants) | 495 | 490
  Potassium, Week 40, n=495, 490 | 0.04 (0.351) | 0.02 (0.334)
  Potassium, Week 48, n=493, 486: number analyzed (Participants) | 493 | 486
  Potassium, Week 48, n=493, 486 | 0.04 (0.315) | 0.03 (0.327)
  Sodium, Week 4, n=326, 520: number analyzed (Participants) | 326 | 520
  Sodium, Week 4, n=326, 520 | 0.4 (2.02) | 0.1 (2.11)
  Sodium, Week 8, n=510, 515: number analyzed (Participants) | 510 | 515
  Sodium, Week 8, n=510, 515 | 0.1 (2.14) | 0.2 (2.02)
  Sodium, Week 16, n=515, 513: number analyzed (Participants) | 515 | 513
  Sodium, Week 16, n=515, 513 | 0.0 (2.00) | -0.1 (2.01)
  Sodium, Week 24, n=505, 503: number analyzed (Participants) | 505 | 503
  Sodium, Week 24, n=505, 503 | -0.2 (2.07) | -0.3 (2.20)
  Sodium, Week 32, n=499, 498: number analyzed (Participants) | 499 | 498
  Sodium, Week 32, n=499, 498 | -0.1 (2.10) | -0.1 (2.21)
  Sodium, Week 40, n=495, 490: number analyzed (Participants) | 495 | 490
  Sodium, Week 40, n=495, 490 | -0.3 (2.09) | -0.2 (2.13)
  Sodium, Week 48, n=493, 486: number analyzed (Participants) | 493 | 486
  Sodium, Week 48, n=493, 486 | -0.4 (2.02) | -0.3 (2.21)
  Urea, Week 4, n=326, 520: number analyzed (Participants) | 326 | 520
  Urea, Week 4, n=326, 520 | 0.24 (1.251) | 0.19 (1.227)
  Urea, Week 8, n=510, 515: number analyzed (Participants) | 510 | 515
  Urea, Week 8, n=510, 515 | 0.07 (1.306) | 0.19 (1.336)
  Urea, Week 16, n=515, 513: number analyzed (Participants) | 515 | 513
  Urea, Week 16, n=515, 513 | 0.07 (1.372) | 0.15 (1.320)
  Urea, Week 24, n=505, 503: number analyzed (Participants) | 505 | 503
  Urea, Week 24, n=505, 503 | 0.06 (1.298) | 0.15 (1.270)
  Urea, Week 32, n=499, 498: number analyzed (Participants) | 499 | 498
  Urea, Week 32, n=499, 498 | 0.11 (1.297) | 0.16 (1.356)
  Urea, Week 40, n=495, 490: number analyzed (Participants) | 495 | 490
  Urea, Week 40, n=495, 490 | 0.18 (1.345) | 0.21 (1.412)
  Urea, Week 48, n=493, 486: number analyzed (Participants) | 493 | 486
  Urea, Week 48, n=493, 486 | 0.13 (1.350) | 0.14 (1.457)

19. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Cholesterol, Glucose, Direct High Density Lipoprotein (HDL) Cholesterol, LDL Cholesterol Calculation and Triglycerides at Week 48
Description: Blood samples were collected for the analysis of clinical chemistry parameters: cholesterol, glucose, direct HDL cholesterol, LDL cholesterol calculation and triglycerides. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and Week 48
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | CAB LA + RPV LA Q8W | CAB LA + RPV LA Q4W
Number analyzed (Participants) | 522 | 523
Millimoles per liter
  Cholesterol, Week 48, n=423, 408: number analyzed (Participants) | 423 | 408
  Cholesterol, Week 48, n=423, 408 | 0.023 (0.742) | 0.075 (0.748)
  Glucose, Week 48, n=478, 470: number analyzed (Participants) | 478 | 470
  Glucose, Week 48, n=478, 470 | 0.16 (0.907) | 0.12 (1.208)
  Direct HDL cholesterol, Week 48, n=423, 408: number analyzed (Participants) | 423 | 408
  Direct HDL cholesterol, Week 48, n=423, 408 | 0.011 (0.292) | -0.000 (0.288)
  LDL cholesterol calculation, Week 48, n=415, 398: number analyzed (Participants) | 415 | 398
  LDL cholesterol calculation, Week 48, n=415, 398 | 0.026 (0.629) | 0.098 (0.585)
  Triglycerides, Week 48, n=423, 408: number analyzed (Participants) | 423 | 408
  Triglycerides, Week 48, n=423, 408 | -0.039 (0.790) | -0.017 (0.880)

20. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter: GFR From Creatinine Adjusted Using Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) Over Time
Description: Blood samples were collected for the analysis of clinical chemistry parameter: GFR from creatinine adjusted using CKD-EPI. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and Weeks 4, 8, 16, 24, 32, 40 and 48
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: milliliters/minute/1.73 square meter
Arm/Group | CAB LA + RPV LA Q8W | CAB LA + RPV LA Q4W
Number analyzed (Participants) | 522 | 523
milliliters/minute/1.73 square meter
  Week 4, n=326, 521: number analyzed (Participants) | 326 | 521
  Week 4, n=326, 521 | -0.8 (9.05) | 0.4 (7.91)
  Week 8, n=508, 514: number analyzed (Participants) | 508 | 514
  Week 8, n=508, 514 | 1.0 (9.07) | 0.4 (8.62)
  Week 16, n=515, 513: number analyzed (Participants) | 515 | 513
  Week 16, n=515, 513 | -0.2 (9.08) | -0.4 (9.01)
  Week 24, n=503, 503: number analyzed (Participants) | 503 | 503
  Week 24, n=503, 503 | -0.7 (9.67) | -1.7 (10.65)
  Week 32, n=499, 498: number analyzed (Participants) | 499 | 498
  Week 32, n=499, 498 | -1.7 (10.12) | -3.0 (10.19)
  Week 40, n=494, 489: number analyzed (Participants) | 494 | 489
  Week 40, n=494, 489 | -1.7 (9.92) | -2.9 (9.95)
  Week 48, n=493, 486: number analyzed (Participants) | 493 | 486
  Week 48, n=493, 486 | -1.9 (9.96) | -3.3 (9.79)

21. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter: Lipase Over Time
Description: Blood samples were collected for the analysis of clinical chemistry parameter: Lipase. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and Weeks 4, 8, 16, 24, 32, 40 and 48
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | CAB LA + RPV LA Q8W | CAB LA + RPV LA Q4W
Number analyzed (Participants) | 522 | 523
Units per liter
  Week 4, n=326, 521: number analyzed (Participants) | 326 | 521
  Week 4, n=326, 521 | 1.7 (28.76) | 1.1 (22.67)
  Week 8, n=510, 514: number analyzed (Participants) | 510 | 514
  Week 8, n=510, 514 | 1.5 (23.82) | 1.4 (24.74)
  Week 16, n=515, 513: number analyzed (Participants) | 515 | 513
  Week 16, n=515, 513 | 2.7 (33.41) | 0.7 (18.82)
  Week 24, n=503, 503: number analyzed (Participants) | 503 | 503
  Week 24, n=503, 503 | 0.7 (19.71) | 2.6 (34.49)
  Week 32, n=499, 498: number analyzed (Participants) | 499 | 498
  Week 32, n=499, 498 | 3.1 (35.20) | -0.5 (21.91)
  Week 40, n=494, 486: number analyzed (Participants) | 494 | 486
  Week 40, n=494, 486 | 1.3 (23.35) | 2.7 (30.95)
  Week 48, n=493, 486: number analyzed (Participants) | 493 | 486
  Week 48, n=493, 486 | 3.2 (53.46) | 2.9 (42.61)

22. Secondary Outcome: Change From Baseline in Hematology Parameters: Basophils, Eosinophils, Leukocytes, Lymphocytes, Monocytes, Neutrophils and Platelets Over Time
Description: Blood samples were collected for the analysis of hematology parameters: basophils, eosinophils, leukocytes, lymphocytes, monocytes, neutrophils and platelets. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and Weeks 4, 8, 16, 24, 32, 40 and 48
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | CAB LA + RPV LA Q8W | CAB LA + RPV LA Q4W
Number analyzed (Participants) | 522 | 523
10^9 cells per liter
  Basophils, Week 4, n=330, 516: number analyzed (Participants) | 330 | 516
  Basophils, Week 4, n=330, 516 | 0.006 (0.02751) | 0.003 (0.02811)
  Basophils, Week 8, n=506, 505: number analyzed (Participants) | 506 | 505
  Basophils, Week 8, n=506, 505 | 0.000 (0.02682) | 0.002 (0.02699)
  Basophils, Week 16, n=508, 507: number analyzed (Participants) | 508 | 507
  Basophils, Week 16, n=508, 507 | -0.000 (0.02651) | 0.001 (0.02929)
  Basophils, Week 24, n=497, 495: number analyzed (Participants) | 497 | 495
  Basophils, Week 24, n=497, 495 | 0.002 (0.02809) | 0.002 (0.02803)
  Basophils, Week 32, n=489, 486: number analyzed (Participants) | 489 | 486
  Basophils, Week 32, n=489, 486 | 0.005 (0.02708) | 0.003 (0.02988)
  Basophils, Week 40, n=479, 472: number analyzed (Participants) | 479 | 472
  Basophils, Week 40, n=479, 472 | 0.004 (0.02716) | 0.004 (0.02772)
  Basophils, Week 48, n=486, 478: number analyzed (Participants) | 486 | 478
  Basophils, Week 48, n=486, 478 | 0.005 (0.02730) | 0.003 (0.02926)
  Eosinophils, Week 4, n=330, 516: number analyzed (Participants) | 330 | 516
  Eosinophils, Week 4, n=330, 516 | 0.031 (0.13775) | 0.015 (0.15112)
  Eosinophils, Week 8, n=506, 505: number analyzed (Participants) | 506 | 505
  Eosinophils, Week 8, n=506, 505 | 0.015 (0.14391) | 0.012 (0.13314)
  Eosinophils, Week 16, n=508, 507: number analyzed (Participants) | 508 | 507
  Eosinophils, Week 16, n=508, 507 | 0.001 (0.13474) | 0.010 (0.13012)
  Eosinophils, Week 24, n=497, 495: number analyzed (Participants) | 497 | 495
  Eosinophils, Week 24, n=497, 495 | 0.001 (0.13607) | 0.009 (0.12836)
  Eosinophils, Week 32, n=489, 486: number analyzed (Participants) | 489 | 486
  Eosinophils, Week 32, n=489, 486 | 0.005 (0.12762) | 0.011 (0.13810)
  Eosinophils, Week 40, n=479, 472: number analyzed (Participants) | 479 | 472
  Eosinophils, Week 40, n=479, 472 | 0.006 (0.13578) | 0.009 (0.12297)
  Eosinophils, Week 48, n=486, 478: number analyzed (Participants) | 486 | 478
  Eosinophils, Week 48, n=486, 478 | 0.001 (0.12444) | 0.002 (0.12646)
  Leukocytes, Week 4, n=331, 520: number analyzed (Participants) | 331 | 520
  Leukocytes, Week 4, n=331, 520 | 0.437 (1.5653) | 0.335 (1.6343)
  Leukocytes, Week 8, n=508, 507: number analyzed (Participants) | 508 | 507
  Leukocytes, Week 8, n=508, 507 | 0.110 (1.5863) | 0.214 (1.6109)
  Leukocytes, Week 16, n=509, 507: number analyzed (Participants) | 509 | 507
  Leukocytes, Week 16, n=509, 507 | 0.050 (1.4281) | 0.139 (1.6384)
  Leukocytes, Week 24, n=499, 497: number analyzed (Participants) | 499 | 497
  Leukocytes, Week 24, n=499, 497 | 0.148 (1.5229) | 0.139 (1.6301)
  Leukocytes, Week 32, n=491, 489: number analyzed (Participants) | 491 | 489
  Leukocytes, Week 32, n=491, 489 | 0.185 (1.5455) | 0.111 (1.6454)
  Leukocytes, Week 40, n=480, 476: number analyzed (Participants) | 480 | 476
  Leukocytes, Week 40, n=480, 476 | 0.177 (1.6601) | 0.100 (1.8042)
  Leukocytes, Week 48, n=488, 478: number analyzed (Participants) | 488 | 478
  Leukocytes, Week 48, n=488, 478 | -0.007 (1.5561) | -0.012 (1.6035)
  Lymphocytes, Week 4, n=330, 516: number analyzed (Participants) | 330 | 516
  Lymphocytes, Week 4, n=330, 516 | 0.187 (0.44013) | 0.063 (0.42683)
  Lymphocytes, Week 8, n=506, 505: number analyzed (Participants) | 506 | 505
  Lymphocytes, Week 8, n=506, 505 | 0.040 (0.39452) | 0.039 (0.44987)
  Lymphocytes, Week 16, n=508, 507: number analyzed (Participants) | 508 | 507
  Lymphocytes, Week 16, n=508, 507 | 0.060 (0.43470) | 0.033 (0.44030)
  Lymphocytes, Week 24, n=497, 495: number analyzed (Participants) | 497 | 495
  Lymphocytes, Week 24, n=497, 495 | 0.081 (0.41863) | 0.061 (0.46240)
  Lymphocytes, Week 32, n=489, 486: number analyzed (Participants) | 489 | 486
  Lymphocytes, Week 32, n=489, 486 | 0.119 (0.46387) | 0.096 (0.45178)
  Lymphocytes, Week 40, n=479, 472: number analyzed (Participants) | 479 | 472
  Lymphocytes, Week 40, n=479, 472 | 0.126 (0.44614) | 0.107 (0.50590)
  Lymphocytes, Week 48, n=486, 478: number analyzed (Participants) | 486 | 478
  Lymphocytes, Week 48, n=486, 478 | 0.063 (0.43255) | 0.049 (0.48991)
  Monocytes, Week 4, n=330, 516: number analyzed (Participants) | 330 | 516
  Monocytes, Week 4, n=330, 516 | 0.051 (0.14208) | 0.021 (0.13359)
  Monocytes, Week 8, n=506, 505: number analyzed (Participants) | 506 | 505
  Monocytes, Week 8, n=506, 505 | 0.003 (0.12080) | 0.003 (0.14270)
  Monocytes, Week 16, n=508, 507: number analyzed (Participants) | 508 | 507
  Monocytes, Week 16, n=508, 507 | -0.002 (0.12804) | -0.007 (0.14361)
  Monocytes, Week 24, n=497, 495: number analyzed (Participants) | 497 | 495
  Monocytes, Week 24, n=497, 495 | 0.019 (0.13460) | 0.020 (0.14458)
  Monocytes, Week 32, n=489, 486: number analyzed (Participants) | 489 | 486
  Monocytes, Week 32, n=489, 486 | 0.048 (0.13969) | 0.039 (0.14531)
  Monocytes, Week 40, n=479, 472: number analyzed (Participants) | 479 | 472
  Monocytes, Week 40, n=479, 472 | 0.060 (0.13570) | 0.060 (0.15692)
  Monocytes, Week 48, n=486, 478: number analyzed (Participants) | 486 | 478
  Monocytes, Week 48, n=486, 478 | 0.030 (0.13329) | 0.033 (0.13116)
  Neutrophils, Week 4, n=330, 516: number analyzed (Participants) | 330 | 516
  Neutrophils, Week 4, n=330, 516 | 0.152 (1.44916) | 0.228 (1.48979)
  Neutrophils, Week 8, n=506, 505: number analyzed (Participants) | 506 | 505
  Neutrophils, Week 8, n=506, 505 | 0.035 (1.49397) | 0.141 (1.48054)
  Neutrophils, Week 16, n=508, 507: number analyzed (Participants) | 508 | 507
  Neutrophils, Week 16, n=508, 507 | -0.018 (1.34384) | 0.082 (1.52187)
  Neutrophils, Week 24, n=497, 495: number analyzed (Participants) | 497 | 495
  Neutrophils, Week 24, n=497, 495 | 0.047 (1.36697) | 0.027 (1.46192)
  Neutrophils, Week 32, n=489, 486: number analyzed (Participants) | 489 | 486
  Neutrophils, Week 32, n=489, 486 | 0.001 (1.43051) | -0.054 (1.53192)
  Neutrophils, Week 40, n=479, 472: number analyzed (Participants) | 479 | 472
  Neutrophils, Week 40, n=479, 472 | -0.021 (1.53092) | -0.090 (1.58850)
  Neutrophils, Week 48, n=486, 478: number analyzed (Participants) | 486 | 478
  Neutrophils, Week 48, n=486, 478 | -0.108 (1.39875) | -0.118 (1.37189)
  Platelets, Week 4, n=329, 518: number analyzed (Participants) | 329 | 518
  Platelets, Week 4, n=329, 518 | 2.09 (32.330) | 5.91 (39.613)
  Platelets, Week 8, n=506, 507: number analyzed (Participants) | 506 | 507
  Platelets, Week 8, n=506, 507 | -0.62 (35.873) | 0.27 (34.345)
  Platelets, Week 16, n=498, 505: number analyzed (Participants) | 498 | 505
  Platelets, Week 16, n=498, 505 | 0.01 (35.207) | -1.70 (34.072)
  Platelets, Week 24, n=496, 496: number analyzed (Participants) | 496 | 496
  Platelets, Week 24, n=496, 496 | 0.26 (36.085) | -2.53 (35.214)
  Platelets, Week 32, n=487, 486: number analyzed (Participants) | 487 | 486
  Platelets, Week 32, n=487, 486 | 1.67 (40.601) | -1.76 (37.490)
  Platelets, Week 40, n=478, 472: number analyzed (Participants) | 478 | 472
  Platelets, Week 40, n=478, 472 | 0.38 (38.636) | 0.32 (38.028)
  Platelets, Week 48, n=489, 474: number analyzed (Participants) | 489 | 474
  Platelets, Week 48, n=489, 474 | 0.06 (39.549) | -1.51 (35.440)

23. Secondary Outcome: Change From Baseline in Hematology Parameter: Erythrocyte Mean Corpuscular Volume (MCV) Over Time
Description: Blood samples were collected for the analysis of hematology parameter: erythrocyte MCV. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and Weeks 4, 8, 16, 24, 32, 40 and 48
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | CAB LA + RPV LA Q8W | CAB LA + RPV LA Q4W
Number analyzed (Participants) | 522 | 523
Femtoliters
  Week 4, n=331, 520: number analyzed (Participants) | 331 | 520
  Week 4, n=331, 520 | -0.32 (2.136) | -0.13 (2.322)
  Week 8, n=509, 510: number analyzed (Participants) | 509 | 510
  Week 8, n=509, 510 | -1.16 (3.270) | -0.84 (3.132)
  Week 16, n=509, 507: number analyzed (Participants) | 509 | 507
  Week 16, n=509, 507 | -1.99 (4.583) | -1.84 (4.370)
  Week 24, n=500, 498: number analyzed (Participants) | 500 | 498
  Week 24, n=500, 498 | -2.46 (5.085) | -2.41 (4.777)
  Week 32, n=491, 491: number analyzed (Participants) | 491 | 491
  Week 32, n=491, 491 | -3.17 (5.005) | -2.75 (4.682)
  Week 40, n=481, 476: number analyzed (Participants) | 481 | 476
  Week 40, n=481, 476 | -3.35 (4.740) | -3.15 (4.578)
  Week 48, n=489, 478: number analyzed (Participants) | 489 | 478
  Week 48, n=489, 478 | -3.28 (5.000) | -3.08 (4.797)

24. Secondary Outcome: Change From Baseline in Hematology Parameter: Erythrocytes Over Time
Description: Blood samples were collected for the analysis of hematology parameter: erythrocytes. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and Weeks 4, 8, 16, 24, 32, 40 and 48
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | CAB LA + RPV LA Q8W | CAB LA + RPV LA Q4W
Number analyzed (Participants) | 522 | 523
10^12 cells per liter
  Week 4, n=331, 520: number analyzed (Participants) | 331 | 520
  Week 4, n=331, 520 | 0.033 (0.2206) | 0.024 (0.2211)
  Week 8, n=509, 510: number analyzed (Participants) | 509 | 510
  Week 8, n=509, 510 | 0.092 (0.2669) | 0.083 (0.2651)
  Week 16, n=509, 507: number analyzed (Participants) | 509 | 507
  Week 16, n=509, 507 | 0.182 (0.3050) | 0.162 (0.3222)
  Week 24, n=500, 498: number analyzed (Participants) | 500 | 498
  Week 24, n=500, 498 | 0.209 (0.3071) | 0.170 (0.3225)
  Week 32, n=491, 491: number analyzed (Participants) | 491 | 491
  Week 32, n=491, 491 | 0.189 (0.3145) | 0.150 (0.3337)
  Week 40, n=481, 476: number analyzed (Participants) | 481 | 476
  Week 40, n=481, 476 | 0.229 (0.3217) | 0.157 (0.3184)
  Week 48, n=489, 478: number analyzed (Participants) | 489 | 478
  Week 48, n=489, 478 | 0.188 (0.3288) | 0.170 (0.3329)

25. Secondary Outcome: Change From Baseline in Hematology Parameter: Hematocrit Over Time
Description: Blood samples were collected for the analysis of hematology parameter: hematocrit. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and Weeks 4, 8, 16, 24, 32, 40 and 48
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | CAB LA + RPV LA Q8W | CAB LA + RPV LA Q4W
Number analyzed (Participants) | 522 | 523
Proportion of red blood cells in blood
  Week 4, n=331, 520: number analyzed (Participants) | 331 | 520
  Week 4, n=331, 520 | 0.002 (0.02088) | 0.002 (0.02202)
  Week 8, n=509, 510: number analyzed (Participants) | 509 | 510
  Week 8, n=509, 510 | 0.004 (0.02274) | 0.004 (0.02362)
  Week 16, n=509, 507: number analyzed (Participants) | 509 | 507
  Week 16, n=509, 507 | 0.008 (0.02290) | 0.007 (0.02485)
  Week 24, n=500, 498: number analyzed (Participants) | 500 | 498
  Week 24, n=500, 498 | 0.008 (0.02219) | 0.004 (0.02413)
  Week 32, n=491, 491: number analyzed (Participants) | 491 | 491
  Week 32, n=491, 491 | 0.003 (0.02352) | 0.001 (0.02469)
  Week 40, n=481, 476: number analyzed (Participants) | 481 | 476
  Week 40, n=481, 476 | 0.006 (0.02323) | 0.000 (0.02378)
  Week 48, n=489, 478: number analyzed (Participants) | 489 | 478
  Week 48, n=489, 478 | 0.003 (0.02414) | 0.001 (0.02565)

26. Secondary Outcome: Change From Baseline in Hematology Parameter: Hemoglobin Over Time
Description: Blood samples were collected for the analysis of hematology parameter: hemoglobin. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and Weeks 4, 8, 16, 24, 32, 40 and 48
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | CAB LA + RPV LA Q8W | CAB LA + RPV LA Q4W
Number analyzed (Participants) | 522 | 523
Grams per liter
  Week 4, n=331, 520: number analyzed (Participants) | 331 | 520
  Week 4, n=331, 520 | 0.08 (6.425) | -0.16 (6.797)
  Week 8, n=509, 510: number analyzed (Participants) | 509 | 510
  Week 8, n=509, 510 | 0.28 (7.028) | -0.05 (7.419)
  Week 16, n=509, 507: number analyzed (Participants) | 509 | 507
  Week 16, n=509, 507 | 0.44 (6.979) | 0.05 (7.531)
  Week 24, n=501, 498: number analyzed (Participants) | 501 | 498
  Week 24, n=501, 498 | 1.48 (7.013) | 0.45 (7.488)
  Week 32, n=491, 491: number analyzed (Participants) | 491 | 491
  Week 32, n=491, 491 | 1.11 (7.633) | 0.05 (8.041)
  Week 40, n=481, 476: number analyzed (Participants) | 481 | 476
  Week 40, n=481, 476 | 1.36 (7.503) | -0.47 (7.788)
  Week 48, n=489, 478: number analyzed (Participants) | 489 | 478
  Week 48, n=489, 478 | -0.13 (7.631) | -0.80 (8.462)

27. Secondary Outcome: Number of Participants With Phenotypic Resistance- Maintenance Phase
Description: Phenotypic resistance (PR) was analyzed in participants who met CVF criteria. PR for following Baseline third agent drugs: Integrase inhibitors(INI): bictegravir (BIC), CAB, dolutegravir (DTG), elvitegravir (EVG), raltegravir(RAL); non-nucleoside reverse transcriptase inhibitors(NNRTI): delavirdine(DLV), efavirenz(EFV), etravirine(ETR), nevirapine(NVP), RPV; nucleoside reverse transcriptase inhibitor (NRTI): lamivudine(3TC), abacavir(ABC), emtricitabine(FTC), tenofovir(TDF), zidovudine(ZDV), stavudine(d4T), didanosine(ddI) and protease inhibitors(PI): atazanavir(ATV), darunavir(DRV), fosamprenavir(FPV), indinavir(IDV), lopinavir(LPV), nelfinavir(NFV), ritonavir(RTV), saquinavir(SQV) and tipranavir (TPV) is presented. Phenotypic susceptibility was defined based on the fold change (FC) value: resistant (FC>clinical higher cutoff or biological cutoff), partially sensitive (FC<=clinical higher cutoff and > clinical lower cutoff), sensitive(FC<=clinical lower cutoff or biological cutoff)
Time Frame: Up to Week 48 analysis
Population: The CVF Population comprised of all participants in ITT-E population who met CVF criteria. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA + RPV LA Q8W | CAB LA + RPV LA Q4W
Number analyzed (Participants) | 8 | 2
Participants
  INI, BIC, resistant, n=6, 2: number analyzed (Participants) | 6 | 2
  INI, BIC, resistant, n=6, 2 | 0 | 0
  INI, BIC, sensitive, n=6, 2: number analyzed (Participants) | 6 | 2
  INI, BIC, sensitive, n=6, 2 | 6 | 2
  INI, CAB, resistant, n=6, 2: number analyzed (Participants) | 6 | 2
  INI, CAB, resistant, n=6, 2 | 3 | 1
  INI, CAB, sensitive, n=6, 2: number analyzed (Participants) | 6 | 2
  INI, CAB, sensitive, n=6, 2 | 3 | 1
  INI, DTG, resistant, n=6, 2: number analyzed (Participants) | 6 | 2
  INI, DTG, resistant, n=6, 2 | 0 | 0
  INI, DTG, partially sensitive, n=6, 2: number analyzed (Participants) | 6 | 2
  INI, DTG, partially sensitive, n=6, 2 | 0 | 0
  INI, DTG, sensitive, n=6, 2: number analyzed (Participants) | 6 | 2
  INI, DTG, sensitive, n=6, 2 | 6 | 2
  INI, EVG, resistant, n=6, 2: number analyzed (Participants) | 6 | 2
  INI, EVG, resistant, n=6, 2 | 4 | 2
  INI, EVG, sensitive, n=6, 2: number analyzed (Participants) | 6 | 2
  INI, EVG, sensitive, n=6, 2 | 2 | 0
  INI, RAL, resistant, n=6, 2: number analyzed (Participants) | 6 | 2
  INI, RAL, resistant, n=6, 2 | 4 | 2
  INI, RAL, sensitive, n=6, 2: number analyzed (Participants) | 6 | 2
  INI, RAL, sensitive, n=6, 2 | 2 | 0
  NNRTI, DLV, resistant, n=7, 2: number analyzed (Participants) | 7 | 2
  NNRTI, DLV, resistant, n=7, 2 | 6 | 2
  NNRTI, DLV, sensitive, n=7, 2: number analyzed (Participants) | 7 | 2
  NNRTI, DLV, sensitive, n=7, 2 | 1 | 0
  NNRTI, EFV, resistant, n=7, 2: number analyzed (Participants) | 7 | 2
  NNRTI, EFV, resistant, n=7, 2 | 5 | 2
  NNRTI, EFV, sensitive, n=7, 2: number analyzed (Participants) | 7 | 2
  NNRTI, EFV, sensitive, n=7, 2 | 2 | 0
  NNRTI, ETR, resistant, n=7, 2: number analyzed (Participants) | 7 | 2
  NNRTI, ETR, resistant, n=7, 2 | 0 | 2
  NNRTI, ETR, partially sensitive, n=7, 2: number analyzed (Participants) | 7 | 2
  NNRTI, ETR, partially sensitive, n=7, 2 | 4 | 0
  NNRTI, ETR, sensitive, n=7, 2: number analyzed (Participants) | 7 | 2
  NNRTI, ETR, sensitive, n=7, 2 | 3 | 0
  NNRTI, NVP, resistant, n=7, 2: number analyzed (Participants) | 7 | 2
  NNRTI, NVP, resistant, n=7, 2 | 6 | 2
  NNRTI, NVP, sensitive, n=7, 2: number analyzed (Participants) | 7 | 2
  NNRTI, NVP, sensitive, n=7, 2 | 1 | 0
  NNRTI, RPV, resistant, n=7, 2: number analyzed (Participants) | 7 | 2
  NNRTI, RPV, resistant, n=7, 2 | 6 | 2
  NNRTI, RPV, sensitive, n=7, 2: number analyzed (Participants) | 7 | 2
  NNRTI, RPV, sensitive, n=7, 2 | 1 | 0
  NRTI, 3TC, resistant, n=7, 2: number analyzed (Participants) | 7 | 2
  NRTI, 3TC, resistant, n=7, 2 | 1 | 1
  NRTI, 3TC, sensitive, n=7, 2: number analyzed (Participants) | 7 | 2
  NRTI, 3TC, sensitive, n=7, 2 | 6 | 1
  NRTI, ABC, resistant, n=7, 2: number analyzed (Participants) | 7 | 2
  NRTI, ABC, resistant, n=7, 2 | 0 | 0
  NRTI, ABC, partially sensitive, n=7, 2: number analyzed (Participants) | 7 | 2
  NRTI, ABC, partially sensitive, n=7, 2 | 0 | 0
  NRTI, ABC, sensitive, n=7, 2: number analyzed (Participants) | 7 | 2
  NRTI, ABC, sensitive, n=7, 2 | 7 | 2
  NRTI, FTC, resistant, n=7, 2: number analyzed (Participants) | 7 | 2
  NRTI, FTC, resistant, n=7, 2 | 1 | 1
  NRTI, FTC, sensitive, n=7, 2: number analyzed (Participants) | 7 | 2
  NRTI, FTC, sensitive, n=7, 2 | 6 | 1
  NRTI, TDF, resistant, n=7, 2: number analyzed (Participants) | 7 | 2
  NRTI, TDF, resistant, n=7, 2 | 0 | 0
  NRTI, TDF, partially sensitive, n=7, 2: number analyzed (Participants) | 7 | 2
  NRTI, TDF, partially sensitive, n=7, 2 | 0 | 1
  NRTI, TDF, sensitive, n=7, 2: number analyzed (Participants) | 7 | 2
  NRTI, TDF, sensitive, n=7, 2 | 7 | 1
  NRTI, ZDV, resistant, n=7, 2: number analyzed (Participants) | 7 | 2
  NRTI, ZDV, resistant, n=7, 2 | 0 | 2
  NRTI, ZDV, sensitive, n=7, 2: number analyzed (Participants) | 7 | 2
  NRTI, ZDV, sensitive, n=7, 2 | 7 | 0
  NRTI, d4T, resistant, n=7, 2: number analyzed (Participants) | 7 | 2
  NRTI, d4T, resistant, n=7, 2 | 0 | 0
  NRTI, d4T, sensitive, n=7, 2: number analyzed (Participants) | 7 | 2
  NRTI, d4T, sensitive, n=7, 2 | 7 | 2
  NRTI, ddI, resistant, n=7, 2: number analyzed (Participants) | 7 | 2
  NRTI, ddI, resistant, n=7, 2 | 0 | 0
  NRTI, ddI, partially sensitive, n=7, 2: number analyzed (Participants) | 7 | 2
  NRTI, ddI, partially sensitive, n=7, 2 | 0 | 0
  NRTI, ddI, sensitive, n=7, 2: number analyzed (Participants) | 7 | 2
  NRTI, ddI, sensitive, n=7, 2 | 7 | 2
  PI, ATV, resistant, n=7, 2: number analyzed (Participants) | 7 | 2
  PI, ATV, resistant, n=7, 2 | 0 | 0
  PI, ATV, sensitive, n=7, 2: number analyzed (Participants) | 7 | 2
  PI, ATV, sensitive, n=7, 2 | 7 | 2
  PI, DRV, resistant, n=7, 2: number analyzed (Participants) | 7 | 2
  PI, DRV, resistant, n=7, 2 | 0 | 0
  PI, DRV, partially sensitive, n=7, 2: number analyzed (Participants) | 7 | 2
  PI, DRV, partially sensitive, n=7, 2 | 0 | 0
  PI, DRV, sensitive, n=7, 2: number analyzed (Participants) | 7 | 2
  PI, DRV, sensitive, n=7, 2 | 7 | 2
  PI, FPV, resistant, n=7, 2: number analyzed (Participants) | 7 | 2
  PI, FPV, resistant, n=7, 2 | 0 | 0
  PI, FPV, partially sensitive, n=7, 2: number analyzed (Participants) | 7 | 2
  PI, FPV, partially sensitive, n=7, 2 | 0 | 0
  PI, FPV, sensitive, n=7, 2: number analyzed (Participants) | 7 | 2
  PI, FPV, sensitive, n=7, 2 | 7 | 2
  PI, IDV, resistant, n=7, 2: number analyzed (Participants) | 7 | 2
  PI, IDV, resistant, n=7, 2 | 0 | 0
  PI, IDV, sensitive, n=7, 2: number analyzed (Participants) | 7 | 2
  PI, IDV, sensitive, n=7, 2 | 7 | 2
  PI, LPV, resistant, n=7, 2: number analyzed (Participants) | 7 | 2
  PI, LPV, resistant, n=7, 2 | 0 | 0
  PI, LPV, partially sensitive, n=7, 2: number analyzed (Participants) | 7 | 2
  PI, LPV, partially sensitive, n=7, 2 | 0 | 0
  PI, LPV, sensitive, n=7, 2: number analyzed (Participants) | 7 | 2
  PI, LPV, sensitive, n=7, 2 | 7 | 2
  PI, NFV, resistant, n=7, 2: number analyzed (Participants) | 7 | 2
  PI, NFV, resistant, n=7, 2 | 0 | 1
  PI, NFV, sensitive, n=7, 2: number analyzed (Participants) | 7 | 2
  PI, NFV, sensitive, n=7, 2 | 7 | 1
  PI, RTV, resistant, n=7, 2: number analyzed (Participants) | 7 | 2
  PI, RTV, resistant, n=7, 2 | 0 | 1
  PI, RTV, sensitive, n=7, 2: number analyzed (Participants) | 7 | 2
  PI, RTV, sensitive, n=7, 2 | 7 | 1
  PI, SQV, resistant, n=7, 2: number analyzed (Participants) | 7 | 2
  PI, SQV, resistant, n=7, 2 | 0 | 0
  PI, SQV, partially sensitive, n=7, 2: number analyzed (Participants) | 7 | 2
  PI, SQV, partially sensitive, n=7, 2 | 0 | 0
  PI, SQV, sensitive, n=7, 2: number analyzed (Participants) | 7 | 2
  PI, SQV, sensitive, n=7, 2 | 7 | 2
  PI, TPV, resistant, n=7, 2: number analyzed (Participants) | 7 | 2
  PI, TPV, resistant, n=7, 2 | 0 | 0
  PI, TPV, partially sensitive, n=7, 2: number analyzed (Participants) | 7 | 2
  PI, TPV, partially sensitive, n=7, 2 | 0 | 0
  PI, TPV, sensitive, n=7, 2: number analyzed (Participants) | 7 | 2
  PI, TPV, sensitive, n=7, 2 | 7 | 2

28. Secondary Outcome: Number of Participants With Genotypic Resistance-Maintenance Phase
Description: Genotypic resistance was analyzed in participants who met confirmed virologic withdrawal criteria. Genotypic Resistance data for the following Baseline third agent drugs, INI: BIC, DTG, EVG, RAL; NNRTI: DLV, EFV, ETR, NVP, RPV; NRTI: 3TC, ABC, FTC, TDF, ZDV, d4T, ddI and PI: ATV, ATV/ritonavir (r), DRV/r, FPV/r, IDV/r, LPV/r, NFV, RTV, SQV/r and TPV/r in participants meeting CVF criteria has been presented.
Time Frame: Up to Week 48 analysis
Population: CVF Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA + RPV LA Q8W | CAB LA + RPV LA Q4W
Number analyzed (Participants) | 8 | 2
Participants
  INI, BIC, resistant, n=6, 2: number analyzed (Participants) | 6 | 2
  INI, BIC, resistant, n=6, 2 | 1 | 0
  INI, BIC, resistance possible, n=6, 2: number analyzed (Participants) | 6 | 2
  INI, BIC, resistance possible, n=6, 2 | 2 | 1
  INI, BIC, sensitive, n=6, 2: number analyzed (Participants) | 6 | 2
  INI, BIC, sensitive, n=6, 2 | 3 | 1
  INI, DTG, resistant, n=6, 2: number analyzed (Participants) | 6 | 2
  INI, DTG, resistant, n=6, 2 | 1 | 0
  INI, DTG, resistance possible, n=6, 2: number analyzed (Participants) | 6 | 2
  INI, DTG, resistance possible, n=6, 2 | 2 | 1
  INI, DTG, sensitive, n=6, 2: number analyzed (Participants) | 6 | 2
  INI, DTG, sensitive, n=6, 2 | 3 | 1
  INI, EVG, resistant, n=6, 2: number analyzed (Participants) | 6 | 2
  INI, EVG, resistant, n=6, 2 | 4 | 2
  INI, EVG, resistance possible, n=6, 2: number analyzed (Participants) | 6 | 2
  INI, EVG, resistance possible, n=6, 2 | 0 | 0
  INI, EVG, sensitive, n=6, 2: number analyzed (Participants) | 6 | 2
  INI, EVG, sensitive, n=6, 2 | 2 | 0
  INI, RAL, resistant, n=6, 2: number analyzed (Participants) | 6 | 2
  INI, RAL, resistant, n=6, 2 | 4 | 2
  INI, RAL, resistance possible, n=6, 2: number analyzed (Participants) | 6 | 2
  INI, RAL, resistance possible, n=6, 2 | 0 | 0
  INI, RAL, sensitive, n=6, 2: number analyzed (Participants) | 6 | 2
  INI, RAL, sensitive, n=6, 2 | 2 | 0
  NNRTI, DLV, resistant, n=8, 2 | 2 | 1
  NNRTI, DLV, resistance possible, n=8, 2 | 2 | 1
  NNRTI, DLV, sensitive, n=8, 2 | 4 | 0
  NNRTI, EFV, resistant, n=8, 2 | 4 | 2
  NNRTI, EFV, resistance possible, n=8, 2 | 2 | 0
  NNRTI, EFV, sensitive, n=8, 2 | 2 | 0
  NNRTI, ETR, resistant, n=8, 2 | 0 | 1
  NNRTI, ETR, resistance possible, n=8, 2 | 2 | 1
  NNRTI, ETR, sensitive, n=8, 2 | 6 | 0
  NNRTI, NVP, resistant, n=8, 2 | 4 | 2
  NNRTI, NVP, resistance possible, n=8, 2 | 2 | 0
  NNRTI, NVP, sensitive, n=8, 2 | 2 | 0
  NNRTI, RPV, resistant, n=8, 2 | 6 | 1
  NNRTI, RPV, resistance possible, n=8, 2 | 0 | 0
  NNRTI, RPV, sensitive, n=8, 2 | 2 | 1
  NRTI, 3TC, resistant, n=8, 2 | 1 | 1
  NRTI, 3TC, resistance possible, n=8, 2 | 0 | 0
  NRTI, 3TC, sensitive, n=8, 2 | 7 | 1
  NRTI, ABC, resistant, n=8, 2 | 0 | 0
  NRTI, ABC, resistance possible, n=8, 2 | 0 | 1
  NRTI, ABC, sensitive, n=8, 2 | 8 | 1
  NRTI, FTC, resistant, n=8, 2 | 1 | 1
  NRTI, FTC, resistance possible, n=8, 2 | 0 | 0
  NRTI, FTC, sensitive, n=8, 2 | 7 | 1
  NRTI, TDF, resistant, n=8, 2 | 0 | 1
  NRTI, TDF, resistance possible, n=8, 2 | 0 | 0
  NRTI, TDF, sensitive, n=8, 2 | 8 | 1
  NRTI, ZDV, resistant, n=8, 2 | 0 | 1
  NRTI, ZDV, resistance possible, n=8, 2 | 0 | 0
  NRTI, ZDV, sensitive, n=8, 2 | 8 | 1
  NRTI, d4T, resistant, n=8, 2 | 0 | 1
  NRTI, d4T, resistance possible, n=8, 2 | 0 | 0
  NRTI, d4T, sensitive, n=8, 2 | 8 | 1
  NRTI, ddI, resistant, n=8, 2 | 0 | 1
  NRTI, ddI, resistance possible, n=8, 2 | 1 | 0
  NRTI, ddI, sensitive, n=8, 2 | 7 | 1
  PI, ATV, resistant, n=8, 2 | 0 | 1
  PI, ATV, resistance possible, n=8, 2 | 0 | 0
  PI, ATV, sensitive, n=8, 2 | 8 | 1
  PI, ATV/r, resistant, n=8, 2 | 0 | 0
  PI, ATV/r, resistance possible, n=8, 2 | 0 | 1
  PI, ATV/r, sensitive, n=8, 2 | 8 | 1
  PI, DRV/r, resistant, n=8, 2 | 0 | 0
  PI, DRV/r, resistance possible, n=8, 2 | 0 | 0
  PI, DRV/r, sensitive, n=8, 2 | 8 | 2
  PI, FPV/r, resistant, n=8, 2 | 0 | 0
  PI, FPV/r, resistance possible, n=8, 2 | 0 | 0
  PI, FPV/r, sensitive, n=8, 2 | 8 | 2
  PI, IDV/r, resistant, n=8, 2 | 0 | 0
  PI, IDV/r, resistance possible, n=8, 2 | 0 | 1
  PI, IDV/r, sensitive, n=8, 2 | 8 | 1
  PI, LPV/r, resistant, n=8, 2 | 0 | 0
  PI, LPV/r, resistance possible, n=8, 2 | 0 | 0
  PI, LPV/r, sensitive, n=8, 2 | 8 | 2
  PI, NFV, resistant, n=8, 2 | 0 | 1
  PI, NFV, resistance possible, n=8, 2 | 0 | 0
  PI, NFV, sensitive, n=8, 2 | 8 | 1
  PI, RTV, resistant, n=8, 2 | 0 | 1
  PI, RTV, resistance possible, n=8, 2 | 0 | 0
  PI, RTV, sensitive, n=8, 2 | 8 | 1
  PI, SQV/r, resistant, n=8, 2 | 0 | 0
  PI, SQV/r, resistance possible, n=8, 2 | 0 | 0
  PI, SQV/r, sensitive, n=8, 2 | 8 | 2
  PI, TPV/r, resistant, n=8, 2 | 0 | 1
  PI, TPV/r, resistance possible, n=8, 2 | 0 | 0
  PI, TPV/r, sensitive, n=8, 2 | 8 | 1

29. Secondary Outcome: Number of Participants With Their Treatment Preference as Assessed Using Preference Questionnaire at Week 48 Without (w/o) Prior Exposure to CAB+RPV-CAB 600 mg LA +RPV 900 mg LA Q8W Arm Only
Description: Participants were administered the preference questionnaire which had 3 questions. For treatment preference, participants were required to provide their response to Question 1, which stated "Based on your experience which HIV treatment do you prefer". The responses included 1) Injectable LA HIV treatment Q4W, 2) Injectable LA HIV Treatment Q8W (only select this answer if you received the 8-week injectable regimen of CAB LA + RPV LA during study), 3) Oral daily HIV treatment and 4) No preference. Oral daily HIV Treatment refers to the oral medication of CAB + RPV subjects received during the oral lead-in period. Number of participants without prior exposure to CAB+RPV who selected each of the responses based on their treatment preference is presented.
Time Frame: Week 48
Population: ITT-E Population. Only those participants with data available at indicated time point is analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA + RPV LA Q8W
Number analyzed (Participants) | 306
Participants
  Injectable LA HIV treatment Q4W | 0
  Injectable LA HIV treatment Q8W | 300
  Oral daily HIV treatment | 4
  No preference | 2

30. Secondary Outcome: Number of Participants With Their Treatment Preference as Assessed Using Preference Questionnaire at Week 48 With >=1 Weeks of Prior Exposure to CAB+RPV-CAB 600 mg LA +RPV 900 mg LA Q8W Arm Only
Description: Participants were administered the preference questionnaire which had 3 questions. For treatment preference, participants were required to provide their response to Question 1, which stated "Based on your experience which HIV treatment do you prefer". The responses included 1) Injectable LA HIV treatment Q4W, 2) Injectable LA HIV Treatment Q8W (only select this answer if you received the 8-week injectable regimen of CAB LA + RPV LA during study), 3) Oral daily HIV treatment and 4) No preference. Oral daily HIV Treatment refers to the oral medication of CAB + RPV subjects received during the oral lead-in period. Number of participants with >=1 weeks of prior exposure to CAB+RPV who selected each of the responses based on their treatment preference is presented.
Time Frame: Week 48
Population: ITT-E Population. Only those participants with data available at indicated time point is analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA + RPV LA Q8W
Number analyzed (Participants) | 191
Participants
  Injectable LA HIV treatment Q4W | 6
  Injectable LA HIV treatment Q8W | 179
  Oral daily HIV treatment | 4
  No preference | 2

31. Secondary Outcome: Number of Participants With Their Treatment Preference as Assessed Using Preference Questionnaire at Week 48-CAB 400 mg LA +RPV 600 mg LA Q4W Arm Only
Description: Participants were administered the preference questionnaire which had 3 questions. For treatment preference, participants were required to provide their response to Question 1, which stated "Based on your experience which HIV treatment do you prefer". The responses included 1) Injectable LA HIV treatment Q4W, 2) Injectable LA HIV Treatment Q8W (only select this answer if you received the 8-week injectable regimen of CAB LA + RPV LA during study), 3) Oral daily HIV treatment and 4) No preference. Oral daily HIV Treatment refers to the oral medication of CAB + RPV participants received during the oral lead-in period. Number of participants who selected each of the responses based on their treatment preference is presented.
Time Frame: Week 48
Population: ITT-E Population. Only those participants with data available at indicated time point is analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA + RPV LA Q4W
Number analyzed (Participants) | 497
Participants
  Injectable LA HIV treatment Q4W | 468
  Injectable LA HIV treatment Q8W | 0
  Oral daily HIV treatment | 16
  No preference | 13

32. Secondary Outcome: Change From Baseline in Life Satisfaction (LISAT) Using HIV/AIDs-targeted Quality of Life (HATQoL) Questionnaire in Participants With or Without Prior Exposure to CAB+RPV
Description: The HATQoL questionnaire was used to assess the health related QoL (HRQoL). It comprises of three dimensions:LISAT, medication worries (MEDWO) and disclosure worries (DISWO). Total imputed value score for LISAT is calculated on a 0-100 scale using the formula: LISAT 100=[100 divided by (20 minus 4)]*(LISAT minus 4). A response of 5 in LISAT score shows satisfaction all of the time and 1 as none of the time. The higher the score, the greater satisfaction to life and the less worry. The transformed dimension score for each domain was summarized and analyzed. Last Observation Carried Forward (LOCF) was used as primary method of analysis. Data for participants without/with prior exposure to CAB+RPV (0 Weeks [without exposure] and >=1 Weeks [with exposure]) has been presented. Baseline value is defined as last available recorded value up to and including the Maintenance treatment start. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1) and Weeks 24 and 48
Population: ITT-E Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | CAB LA + RPV LA Q8W | CAB LA + RPV LA Q4W
Number analyzed (Participants) | 522 | 523
Scores on a scale
  Without exposure, Week 24, n=318, 324: number analyzed (Participants) | 318 | 324
  Without exposure, Week 24, n=318, 324 | 1.5 (14.87) | -0.5 (18.00)
  Without exposure, Week 48, n=319, 324: number analyzed (Participants) | 319 | 324
  Without exposure, Week 48, n=319, 324 | -0.8 (15.24) | 0.6 (17.51)
  With exposure, Week 24, n=192, 194: number analyzed (Participants) | 192 | 194
  With exposure, Week 24, n=192, 194 | -0.8 (14.31) | 0.8 (13.73)
  With exposure, Week 48, n=192, 194: number analyzed (Participants) | 192 | 194
  With exposure, Week 48, n=192, 194 | 0.3 (14.03) | -1.3 (14.50)

33. Secondary Outcome: Change From Baseline in HIV Medication, MEDWO Using HATQoL Questionnaire in Participants With or Without Prior Exposure to CAB+RPV
Description: The HATQoL questionnaire was used to assess the HRQoL. It comprises of three dimensions:LISAT, MEDWO and DISWO. The total imputed value score for MEDWO is calculated on a 0-100 scale using the formula: MEDWO 100=[100 divided by (25 minus 5)]*(MEDWO minus 5). A response of 1 in MEDWO score shows medication worries all of the time and 5 as none of the time. The higher the score, the greater satisfaction to life and the less worry. The transformed dimension score for each domain was summarized and analyzed. LOCF was used as primary method of analysis. Participants without/with prior exposure to CAB+RPV (0 Weeks [without exposure] and >=1 Weeks [with exposure]) has been presented. Baseline value is defined as last available recorded value up to and including the Maintenance treatment start. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1) and Weeks 24 and 48
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | CAB LA + RPV LA Q8W | CAB LA + RPV LA Q4W
Number analyzed (Participants) | 522 | 523
Scores on a scale
  Without exposure, Week 24, n=318, 324: number analyzed (Participants) | 318 | 324
  Without exposure, Week 24, n=318, 324 | 2.7 (16.53) | 2.6 (15.61)
  Without exposure, Week 48, n=319, 324: number analyzed (Participants) | 319 | 324
  Without exposure, Week 48, n=319, 324 | 3.0 (15.87) | 1.9 (15.97)
  With exposure, Week 24, n=192, 194: number analyzed (Participants) | 192 | 194
  With exposure, Week 24, n=192, 194 | 0.7 (10.57) | 1.7 (14.86)
  With exposure, Week 48, n=192, 194: number analyzed (Participants) | 192 | 194
  With exposure, Week 48, n=192, 194 | 1.3 (8.82) | 1.3 (17.95)

34. Secondary Outcome: Change From Baseline in DISWO Using HATQoL Questionnaire in Participants With or Without Prior Exposure to CAB+RPV
Description: The HATQoL questionnaire was used to assess the HRQoL. It comprises of three dimensions:LISAT, MEDWO and DISWO. The total imputed value score for DISWO is calculated on a 0-100 scale using the formula: DISWO 100=[100 divided by (25 minus 5)]*(DISWO minus 5). A response of 1 in DISWO score shows disclosure worries all of the time and 5 as none of the time. The higher the score, the greater satisfaction to life and the less worry. The transformed dimension score for each domain was summarized and analyzed. LOCF was used as primary method of analysis. Participants without/with prior exposure to CAB+RPV (0 Weeks [without exposure] and >=1 Weeks [with exposure]) has been presented. Baseline value is defined as last available recorded value up to and including the Maintenance treatment start. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1) and Weeks 24 and 48
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | CAB LA + RPV LA Q8W | CAB LA + RPV LA Q4W
Number analyzed (Participants) | 522 | 523
Scores on a scale
  Without exposure, Week 24, n=317, 324: number analyzed (Participants) | 317 | 324
  Without exposure, Week 24, n=317, 324 | 1.4 (25.58) | 1.2 (23.18)
  Without exposure, Week 48, n=318, 324: number analyzed (Participants) | 318 | 324
  Without exposure, Week 48, n=318, 324 | -0.5 (28.14) | -0.5 (23.86)
  With exposure, Week 24, n=192, 194: number analyzed (Participants) | 192 | 194
  With exposure, Week 24, n=192, 194 | 0.9 (21.13) | 1.8 (24.20)
  With exposure, Week 48, n=192, 194: number analyzed (Participants) | 192 | 194
  With exposure, Week 48, n=192, 194 | -0.6 (24.11) | 1.5 (26.84)

35. Secondary Outcome: Change From Baseline in Total Treatment Satisfaction Score Using HIV Treatment Satisfaction Status Questionnaire (HIVTSQs) at Weeks 24 and 48
Description: The HIVTSQs treatment satisfaction questionnaire comprises of 1-12 questions and the total treatment satisfaction score is computed with items 1-11 and summed to produce a score with a possible range of 0 to 66. Higher scores represent greater treatment satisfaction as compared to the past few weeks. LOCF was used as primary method of analysis. Participants without/with prior exposure to CAB+RPV (0 Weeks [without exposure] and >=1 Weeks [with exposure]) has been presented. Baseline value is defined as last available recorded value up to and including the Maintenance treatment start. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1) and Weeks 24 and 48
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | CAB LA + RPV LA Q8W | CAB LA + RPV LA Q4W
Number analyzed (Participants) | 522 | 523
Scores on a scale
  Without exposure, Week 24, n=319, 323: number analyzed (Participants) | 319 | 323
  Without exposure, Week 24, n=319, 323 | 4.63 (9.818) | 4.44 (9.709)
  Without exposure, Week 48, n=319, 323: number analyzed (Participants) | 319 | 323
  Without exposure, Week 48, n=319, 323 | 4.42 (10.351) | 3.55 (10.224)
  With exposure, Week 24, n=191, 193: number analyzed (Participants) | 191 | 193
  With exposure, Week 24, n=191, 193 | 0.55 (5.050) | 0.55 (5.347)
  With exposure, Week 48, n=191, 194: number analyzed (Participants) | 191 | 194
  With exposure, Week 48, n=191, 194 | 0.40 (5.242) | -0.01 (6.521)

36. Secondary Outcome: Change From Baseline in Individual Item Scores Using HIVTSQs at Weeks 24 and 48
Description: HIVTSQs is a 12 item questionnaire. The individual item scores on HIVTSQs scale are rated as 6 (very satisfied, convenient, flexible, etc.) to 0 (very dissatisfied, inconvenient, inflexible, etc.). Higher scores represent greater satisfaction with each aspect of treatment. LOCF was used as primary method of analysis. Participants without/with prior exposure to CAB+RPV (0 Weeks [without exposure] and >=1 Weeks [with exposure]) has been presented. Baseline value is defined as last available recorded value up to and including the Maintenance treatment start. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1) and Weeks 24 and 48
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | CAB LA + RPV LA Q8W | CAB LA + RPV LA Q4W
Number analyzed (Participants) | 522 | 523
Scores on a scale
  Item 1, Without exposure, Week 24, n=319, 323: number analyzed (Participants) | 319 | 323
  Item 1, Without exposure, Week 24, n=319, 323 | 0.3 (1.19) | 0.3 (1.18)
  Item 1, Without exposure, Week 48, n=319, 323: number analyzed (Participants) | 319 | 323
  Item 1, Without exposure, Week 48, n=319, 323 | 0.3 (1.23) | 0.2 (1.27)
  Item 1, With exposure, Week 24, n=191, 193: number analyzed (Participants) | 191 | 193
  Item 1, With exposure, Week 24, n=191, 193 | 0.1 (0.77) | 0.0 (0.78)
  Item 1, With exposure, Week 48, n=191, 194: number analyzed (Participants) | 191 | 194
  Item 1, With exposure, Week 48, n=191, 194 | 0.1 (0.81) | 0.0 (0.90)
  Item 2, Without exposure, Week 24, n=319, 323: number analyzed (Participants) | 319 | 323
  Item 2, Without exposure, Week 24, n=319, 323 | 0.0 (0.73) | 0.1 (0.67)
  Item 2, Without exposure, Week 48, n=319, 323: number analyzed (Participants) | 319 | 323
  Item 2, Without exposure, Week 48, n=319, 323 | 0.0 (0.78) | 0.0 (0.65)
  Item 2, With exposure, Week 24, n=191, 193: number analyzed (Participants) | 191 | 193
  Item 2, With exposure, Week 24, n=191, 193 | 0.0 (0.42) | 0.1 (0.61)
  Item 2, With exposure, Week 48, n=191, 194: number analyzed (Participants) | 191 | 194
  Item 2, With exposure, Week 48, n=191, 194 | 0.0 (0.49) | 0.1 (0.63)
  Item 3, Without exposure, Week 24, n=319, 323: number analyzed (Participants) | 319 | 323
  Item 3, Without exposure, Week 24, n=319, 323 | 0.0 (1.42) | 0.0 (1.49)
  Item 3, Without exposure, Week 48, n=319, 323: number analyzed (Participants) | 319 | 323
  Item 3, Without exposure, Week 48, n=319, 323 | 0.0 (1.45) | 0.0 (1.48)
  Item 3, With exposure, Week 24, n=191, 193: number analyzed (Participants) | 191 | 193
  Item 3, With exposure, Week 24, n=191, 193 | 0.0 (0.82) | 0.1 (1.03)
  Item 3, With exposure, Week 48, n=191, 194: number analyzed (Participants) | 191 | 194
  Item 3, With exposure, Week 48, n=191, 194 | 0.0 (1.05) | 0.0 (1.20)
  Item 4, Without exposure, Week 24, n=319, 323: number analyzed (Participants) | 319 | 323
  Item 4, Without exposure, Week 24, n=319, 323 | 0.3 (1.05) | 0.3 (1.28)
  Item 4, Without exposure, Week 48, n=319, 323: number analyzed (Participants) | 319 | 323
  Item 4, Without exposure, Week 48, n=319, 323 | 0.2 (1.20) | 0.2 (1.28)
  Item 4, With exposure, Week 24, n=191, 193: number analyzed (Participants) | 191 | 193
  Item 4, With exposure, Week 24, n=191, 193 | 0.1 (0.73) | 0.0 (0.80)
  Item 4, With exposure, Week 48, n=191, 194: number analyzed (Participants) | 191 | 194
  Item 4, With exposure, Week 48, n=191, 194 | 0.1 (0.73) | 0.0 (0.98)
  Item 5, Without exposure, Week 24, n=319, 323: number analyzed (Participants) | 319 | 323
  Item 5, Without exposure, Week 24, n=319, 323 | 0.7 (1.41) | 0.6 (1.37)
  Item 5, Without exposure, Week 48, n=319, 323: number analyzed (Participants) | 319 | 323
  Item 5, Without exposure, Week 48, n=319, 323 | 0.7 (1.36) | 0.5 (1.42)
  Item 5, With exposure, Week 24, n=191, 193: number analyzed (Participants) | 191 | 193
  Item 5, With exposure, Week 24, n=191, 193 | 0.0 (0.58) | 0.1 (0.72)
  Item 5, With exposure, Week 48, n=191, 194: number analyzed (Participants) | 191 | 194
  Item 5, With exposure, Week 48, n=191, 194 | 0.0 (0.69) | 0.0 (0.88)
  Item 6, Without exposure, Week 24, n=319, 323: number analyzed (Participants) | 319 | 323
  Item 6, Without exposure, Week 24, n=319, 323 | 0.9 (1.72) | 0.8 (1.71)
  Item 6, Without exposure, Week 48, n=319, 323: number analyzed (Participants) | 319 | 323
  Item 6, Without exposure, Week 48, n=319, 323 | 0.8 (1.71) | 0.8 (1.80)
  Item 6, With exposure, Week 24, n=191, 193: number analyzed (Participants) | 191 | 193
  Item 6, With exposure, Week 24, n=191, 193 | 0.2 (0.96) | 0.1 (0.90)
  Item 6, With exposure, Week 48, n=191, 194: number analyzed (Participants) | 191 | 194
  Item 6, With exposure, Week 48, n=191, 194 | 0.1 (1.13) | -0.1 (1.12)
  Item 7, Without exposure, Week 24, n=319, 323: number analyzed (Participants) | 319 | 323
  Item 7, Without exposure, Week 24, n=319, 323 | 0.3 (0.78) | 0.2 (0.98)
  Item 7, Without exposure, Week 48, n=319, 323: number analyzed (Participants) | 319 | 323
  Item 7, Without exposure, Week 48, n=319, 323 | 0.2 (0.94) | 0.2 (0.92)
  Item 7, With exposure, Week 24, n=191, 193: number analyzed (Participants) | 191 | 193
  Item 7, With exposure, Week 24, n=191, 193 | 0.0 (0.55) | 0.0 (0.70)
  Item 7, With exposure, Week 48, n=191, 194: number analyzed (Participants) | 191 | 194
  Item 7, With exposure, Week 48, n=191, 194 | 0.1 (0.73) | 0.1 (0.69)
  Item 8, Without exposure, Week 24, n=318, 322: number analyzed (Participants) | 318 | 322
  Item 8, Without exposure, Week 24, n=318, 322 | 0.5 (1.31) | 0.6 (1.30)
  Item 8, Without exposure, Week 48, n=319, 323: number analyzed (Participants) | 319 | 323
  Item 8, Without exposure, Week 48, n=319, 323 | 0.5 (1.31) | 0.5 (1.41)
  Item 8, With exposure, Week 24, n=191, 194: number analyzed (Participants) | 191 | 194
  Item 8, With exposure, Week 24, n=191, 194 | 0.1 (0.61) | 0.1 (0.58)
  Item 8, With exposure, Week 48, n=191, 194: number analyzed (Participants) | 191 | 194
  Item 8, With exposure, Week 48, n=191, 194 | 0.0 (0.64) | 0.0 (0.80)
  Item 9, Without exposure, Week 24, n=319, 322: number analyzed (Participants) | 319 | 322
  Item 9, Without exposure, Week 24, n=319, 322 | 0.4 (1.16) | 0.4 (1.30)
  Item 9, Without exposure, Week 48, n=319, 323: number analyzed (Participants) | 319 | 323
  Item 9, Without exposure, Week 48, n=319, 323 | 0.4 (1.23) | 0.3 (1.36)
  Item 9, With exposure, Week 24, n=191, 194: number analyzed (Participants) | 191 | 194
  Item 9, With exposure, Week 24, n=191, 194 | 0.0 (0.52) | 0.0 (0.72)
  Item 9, With exposure, Week 48, n=191, 194: number analyzed (Participants) | 191 | 194
  Item 9, With exposure, Week 48, n=191, 194 | 0.1 (0.55) | 0.0 (0.85)
  Item 10, Without exposure, Week 24, n=319, 322: number analyzed (Participants) | 319 | 322
  Item 10, Without exposure, Week 24, n=319, 322 | 0.8 (1.44) | 0.9 (1.50)
  Item 10, Without exposure, Week 48, n=319, 323: number analyzed (Participants) | 319 | 323
  Item 10, Without exposure, Week 48, n=319, 323 | 0.8 (1.52) | 0.7 (1.63)
  Item 10, With exposure, Week 24, n=191, 194: number analyzed (Participants) | 191 | 194
  Item 10, With exposure, Week 24, n=191, 194 | 0.0 (0.78) | 0.0 (0.67)
  Item 10, With exposure, Week 48, n=191, 194: number analyzed (Participants) | 191 | 194
  Item 10, With exposure, Week 48, n=191, 194 | 0.0 (0.79) | 0.0 (0.77)
  Item 11, Without exposure, Week 24, n=319, 322: number analyzed (Participants) | 319 | 322
  Item 11, Without exposure, Week 24, n=319, 322 | 0.4 (1.22) | 0.4 (1.25)
  Item 11, Without exposure, Week 48, n=319, 323: number analyzed (Participants) | 319 | 323
  Item 11, Without exposure, Week 48, n=319, 323 | 0.4 (1.26) | 0.3 (1.31)
  Item 11, With exposure, Week 24, n=191, 194: number analyzed (Participants) | 191 | 194
  Item 11, With exposure, Week 24, n=191, 194 | 0.0 (0.73) | 0.1 (0.65)
  Item 11, With exposure, Week 48, n=191, 194: number analyzed (Participants) | 191 | 194
  Item 11, With exposure, Week 48, n=191, 194 | 0.0 (0.62) | -0.1 (0.84)
  Item 12, Without exposure, Week 24, n=319, 322: number analyzed (Participants) | 319 | 322
  Item 12, Without exposure, Week 24, n=319, 322 | -0.4 (1.46) | -0.4 (1.48)
  Item 12, Without exposure, Week 48, n=319, 323: number analyzed (Participants) | 319 | 323
  Item 12, Without exposure, Week 48, n=319, 323 | -0.3 (1.46) | -0.5 (1.57)
  Item 12, With exposure, Week 24, n=191, 194: number analyzed (Participants) | 191 | 194
  Item 12, With exposure, Week 24, n=191, 194 | -0.1 (0.92) | 0.0 (0.92)
  Item 12, With exposure, Week 48, n=191, 194: number analyzed (Participants) | 191 | 194
  Item 12, With exposure, Week 48, n=191, 194 | -0.1 (1.08) | 0.0 (1.02)

37. Secondary Outcome: Total Treatment Satisfaction Change Score Using HIV Treatment Satisfaction Change Questionnaire (HIVTSQc) at Week 48
Description: The HIVTSQc is a 1-12 items questionnaire. Each item is scored -3 to 3. Total treatment satisfaction change score is computed using items 1 to 11 and are summed to produce a score with a possible range of -33 to 33. Higher the score, greater the improvement in satisfaction with treatment; the lower the score, the greater the deterioration in satisfaction with treatment. A score of 0 represented no change. LOCF was used as primary method of analysis. Total treatment satisfaction change score for participants who entered the current study from Q4W arm of ATLAS (NCT number: NCT02951052) and from either standard of care (SOC) arms of ATLAS or the new SOC participants) has been presented.
Time Frame: Week 48
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | CAB LA + RPV LA Q8W | CAB LA + RPV LA Q4W
Number analyzed (Participants) | 522 | 523
Scores on a scale
  Q4W ATLAS, n=124, 125: number analyzed (Participants) | 124 | 125
  Q4W ATLAS, n=124, 125 | 29.1 (6.72) | 24.7 (12.33)
  SOC, n=380, 382: number analyzed (Participants) | 380 | 382
  SOC, n=380, 382 | 28.9 (7.68) | 27.3 (9.50)

38. Secondary Outcome: Change From Week 8 in Dimension Scores Using Perception of Injection (PIN) Questionnaire.
Description: The PIN questionnaire explores bother of pain at injection site and injection site reactions (ISR), anxiety before and after injection, willingness to receive an HIV injectable treatment the following visit and satisfaction with mode of treatment administration of individuals receiving injection and perceptions of individuals associated with receiving injections. This measure contains 21 items that measure pain at injection site, local site reactions, impact on functioning and willingness to pursue injectable treatment outside of a clinical trial. Scores range from 1 to 5, and questions are phrased in such a way as to ensure that 1 always equated with the most favourable perception of vaccination, and 5 most unfavourable. Dimension scores include bother from ISR, leg movement, sleep and acceptability. Score of a domain is calculated as mean of all items within the domain. Higher scores represent worse perception of injection. LOCF was used as primary method of analysis.
Time Frame: Week 8 and Weeks 24 and 48
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | CAB LA + RPV LA Q8W | CAB LA + RPV LA Q4W
Number analyzed (Participants) | 522 | 523
Scores on a scale
  Bother of ISRs, Week 24, n=515, 515: number analyzed (Participants) | 515 | 515
  Bother of ISRs, Week 24, n=515, 515 | -0.00 (0.459) | -0.01 (0.509)
  Bother of ISRs, Week 48, n=515, 515: number analyzed (Participants) | 515 | 515
  Bother of ISRs, Week 48, n=515, 515 | -0.00 (0.531) | 0.01 (0.543)
  Leg Movement, Week 24, n=515, 514: number analyzed (Participants) | 515 | 514
  Leg Movement, Week 24, n=515, 514 | -0.11 (0.804) | -0.23 (0.809)
  Leg Movement, Week 48, n=515, 514: number analyzed (Participants) | 515 | 514
  Leg Movement, Week 48, n=515, 514 | -0.12 (0.818) | -0.24 (0.789)
  Sleep, Week 24, n=515, 514: number analyzed (Participants) | 515 | 514
  Sleep, Week 24, n=515, 514 | -0.00 (0.772) | -0.20 (0.793)
  Sleep, Week 48, n=515, 514: number analyzed (Participants) | 515 | 514
  Sleep, Week 48, n=515, 514 | -0.03 (0.814) | -0.18 (0.804)
  Acceptance, Week 24, n=514, 515: number analyzed (Participants) | 514 | 515
  Acceptance, Week 24, n=514, 515 | -0.13 (0.813) | -0.13 (0.837)
  Acceptance, Week 48, n=514, 515: number analyzed (Participants) | 514 | 515
  Acceptance, Week 48, n=514, 515 | -0.18 (0.829) | -0.13 (0.880)

39. Secondary Outcome: Change From Week 8 in Individual Item Scores (Anxiety Before, Pain, Satisfaction, Anxiety After and Willingness) Using Perception of Injection (PIN) Questionnaire.
Description: The PIN questionnaire explores the bother of pain at the injection site and ISRs, anxiety before and after injection, willingness to receive an HIV injectable treatment the following visit and satisfaction with the mode of treatment administration of individuals receiving injection and perceptions of individuals associated with receiving injections. This measure contains 21 items that measure pain at injection site, local site reactions, impact on functioning and willingness to pursue injectable treatment outside of a clinical trial. The items in the scale are rated on a 5-point scale ranging from 1(very dissatisfied, extremely, etc.) to 5 (very satisfied, not at all, etc.). Lower scores represent worse perception of injection. LOCF was used as primary method of analysis.
Time Frame: Week 8 and Weeks 24 and 48
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | CAB LA + RPV LA Q8W | CAB LA + RPV LA Q4W
Number analyzed (Participants) | 522 | 523
Scores on a scale
  Anxiety before, Week 24, n=515, 515: number analyzed (Participants) | 515 | 515
  Anxiety before, Week 24, n=515, 515 | 0.0 (0.83) | -0.1 (0.85)
  Anxiety before, Week 48, n=515, 515: number analyzed (Participants) | 515 | 515
  Anxiety before, Week 48, n=515, 515 | -0.1 (0.82) | -0.1 (0.85)
  Pain, Week 24, n=515, 515: number analyzed (Participants) | 515 | 515
  Pain, Week 24, n=515, 515 | 0.1 (0.83) | 0.1 (0.84)
  Pain, Week 48, n=515, 515: number analyzed (Participants) | 515 | 515
  Pain, Week 48, n=515, 515 | 0.0 (0.85) | 0.0 (0.84)
  Satisfaction, Week 24, n=514, 515: number analyzed (Participants) | 514 | 515
  Satisfaction, Week 24, n=514, 515 | 0.1 (0.77) | -0.0 (0.77)
  Satisfaction, Week 48, n=514, 515: number analyzed (Participants) | 514 | 515
  Satisfaction, Week 48, n=514, 515 | -0.0 (0.77) | -0.0 (0.84)
  Anxiety after, Week 24, n=514, 515: number analyzed (Participants) | 514 | 515
  Anxiety after, Week 24, n=514, 515 | -0.0 (0.76) | 0.0 (0.83)
  Anxiety after, Week 48, n=514, 515: number analyzed (Participants) | 514 | 515
  Anxiety after, Week 48, n=514, 515 | -0.1 (0.79) | -0.1 (0.89)
  Willingness, Week 24, n=514, 514: number analyzed (Participants) | 514 | 514
  Willingness, Week 24, n=514, 514 | -0.1 (0.55) | -0.1 (0.65)
  Willingness, Week 48, n=514, 514: number analyzed (Participants) | 514 | 514
  Willingness, Week 48, n=514, 514 | -0.0 (0.66) | -0.1 (0.72)

40. Secondary Outcome: Change From Baseline in Treatment Acceptance a Using "General Acceptance" Dimension of the Chronic Treatment Acceptance (ACCEPT) Questionnaire in Participants With or Without Prior Exposure to CAB+RPV
Description: The ACCEPT questionnaire is a generic medication acceptance measure assessing how participants weigh advantages and disadvantages of long-term medication.The questionnaire consists of 25 items that capture six dimensions.3 questions that focus on general acceptance of study medication were analyzed.Items on the scale are rated as 1-5 scores:1:not at all acceptable,2:not very acceptable,3:somewhat acceptable, 4:totally acceptable and 5:I don't know.Total score of the dimension is calculated as the mean of recoded items of the dimension and then linearly transformed to be on a scale from 0 to 100:Total Score=(mean of the recoded items in the dimension minus1)divided by2*100. LOCF was used as primary method of analysis. Data for participants without or with prior exposure has been presented. Baseline value is defined as last available value up to and including the Maintenance treatment. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1) and Weeks 24 and 48
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | CAB LA + RPV LA Q8W | CAB LA + RPV LA Q4W
Number analyzed (Participants) | 522 | 523
Scores on a scale
  Without exposure, Week 24, n=319, 323: number analyzed (Participants) | 319 | 323
  Without exposure, Week 24, n=319, 323 | 6.0 (27.96) | 4.0 (33.53)
  Without exposure, Week 48, n=319, 324: number analyzed (Participants) | 319 | 324
  Without exposure, Week 48, n=319, 324 | 6.9 (30.96) | 5.6 (31.77)
  With exposure, Week 24, n=192, 194: number analyzed (Participants) | 192 | 194
  With exposure, Week 24, n=192, 194 | 0.3 (21.37) | -1.7 (21.79)
  With exposure, Week 48, n=192, 194: number analyzed (Participants) | 192 | 194
  With exposure, Week 48, n=192, 194 | -0.1 (24.92) | -2.7 (24.25)

41. Secondary Outcome: Plasma Trough Concentration (Ctrough) for CAB LA Evaluable
Description: Blood samples were collected at indicated time points for pharmacokinetic (PK) analysis of CAB LA. PK Population comprises of all participants who received CAB and / or RPV and underwent PK sampling during the study and provide at least 1 non-missing CAB and / or RPV plasma concentration value (Non-quantifiable [NQ] values will be considered as non-missing values).
Time Frame: Pre-dose at Weeks 4, 8, 16, 24, 32, 40 and 48
Population: PK Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Geometric Mean (95% Confidence Interval); unit: Micrograms per milliliter
Groups:
- CAB LA Q8W: Participants in this arm received 2 x 3ml CAB LA injections at week 4b and 2 x 3 ml CAB LA injections Q8W thereafter
- CAB LA Q4W: Participants in this arm received 2 x 3ml CAB LA injections at week 4b and 2 x 2 ml CAB LA injections Q4W thereafter
Arm/Group | CAB LA Q8W | CAB LA Q4W
Number analyzed (Participants) | 521 | 521
Micrograms per milliliter
  Pre-dose, Week 4, n=314, 513: number analyzed (Participants) | 314 | 513
  Pre-dose, Week 4, n=314, 513 | 5.1543 [4.8702 to 5.4550] | 4.0285 [3.8303 to 4.2369]
  Pre-dose, Week 8, n=516, 513: number analyzed (Participants) | 516 | 513
  Pre-dose, Week 8, n=516, 513 | 1.7938 [1.7007 to 1.8920] | 1.9011 [1.7965 to 2.0119]
  Pre-dose, Week 16, n=512, 514: number analyzed (Participants) | 512 | 514
  Pre-dose, Week 16, n=512, 514 | 1.5983 [1.5223 to 1.6781] | 2.3358 [2.2436 to 2.4317]
  Pre-dose, Week 24, n=506, 510: number analyzed (Participants) | 506 | 510
  Pre-dose, Week 24, n=506, 510 | 1.5955 [1.5203 to 1.6744] | 2.5795 [2.4826 to 2.6802]
  Pre-dose, Week 32, n=499, 498: number analyzed (Participants) | 499 | 498
  Pre-dose, Week 32, n=499, 498 | 1.7414 [1.6612 to 1.8254] | 2.8529 [2.7408 to 2.9696]
  Pre-dose, Week 40, n=496, 497: number analyzed (Participants) | 496 | 497
  Pre-dose, Week 40, n=496, 497 | 1.7873 [1.7058 to 1.8727] | 2.9739 [2.8713 to 3.0801]
  Pre-dose, Week 48, n=494, 486: number analyzed (Participants) | 494 | 486
  Pre-dose, Week 48, n=494, 486 | 1.6747 [1.6033 to 1.7493] | 2.7449 [2.6492 to 2.8441]

42. Secondary Outcome: Plasma Ctrough for RPV LA Evaluable
Description: Blood samples were collected at indicated time points for PK analysis of RPV LA.
Time Frame: Pre-dose at Weeks 4, 8, 16, 24, 32, 40 and 48
Population: as for outcome 41
Measure: Geometric Mean (95% Confidence Interval); unit: Nanograms per milliliters
Groups:
- RPV LA Q8W: Participants in this arm received 2 x 3ml RPV LA injections at week 4b and 2 x 3 ml RPV LA injections Q8W thereafter
- RPV LA Q4W: Participants in this arm received 2 x 3ml RPV LA injections at week 4b and 2 x 2 ml RPV LA injections Q4W thereafter
Arm/Group | RPV LA Q8W | RPV LA Q4W
Number analyzed (Participants) | 521 | 521
Nanograms per milliliters
  Pre-dose, Week 4, n=315, 514: number analyzed (Participants) | 315 | 514
  Pre-dose, Week 4, n=315, 514 | 78.05 [73.32 to 83.09] | 78.60 [75.03 to 82.35]
  Pre-dose, Week 8, n=515, 512: number analyzed (Participants) | 515 | 512
  Pre-dose, Week 8, n=515, 512 | 56.35 [53.73 to 59.09] | 57.95 [55.09 to 60.96]
  Pre-dose, Week 16, n=512, 513: number analyzed (Participants) | 512 | 513
  Pre-dose, Week 16, n=512, 513 | 54.84 [52.55 to 57.22] | 68.12 [65.15 to 71.23]
  Pre-dose, Week 24, n=506, 509: number analyzed (Participants) | 506 | 509
  Pre-dose, Week 24, n=506, 509 | 57.16 [54.77 to 59.66] | 75.76 [72.64 to 79.02]
  Pre-dose, Week 32, n=498, 498: number analyzed (Participants) | 498 | 498
  Pre-dose, Week 32, n=498, 498 | 62.07 [59.54 to 64.71] | 85.76 [82.35 to 89.30]
  Pre-dose, Week 40, n=497, 497: number analyzed (Participants) | 497 | 497
  Pre-dose, Week 40, n=497, 497 | 67.22 [64.58 to 69.97] | 89.49 [86.22 to 92.88]
  Pre-dose, Week 48, n=495, 488: number analyzed (Participants) | 495 | 488
  Pre-dose, Week 48, n=495, 488 | 72.29 [69.50 to 75.19] | 97.22 [93.49 to 101.09]

43. Secondary Outcome: Area Under the Curve (AUC) for CAB LA
Description: Blood samples were collected at indicated time points to analyze concentration in plasma for CAB LA. Participants who transitioned from ATLAS (201585 - NCT02951052) into this ATLAS-2M (207966) study had been treated with CAB + RPV for at least one year, were approaching steady state exposures, and were therefore excluded in order to focus the population analysis on those without prior exposure.
Time Frame: Predose at Weeks 4, 8, 13, 24, 32, 40, 48; 1 Week post-dose at Week 9 and 41
Population: PK Population. Only those participants with data available at specified time points has been analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Micrograms*hours per milliliter
Arm/Group | CAB LA Q8W | CAB LA Q4W
Number analyzed (Participants) | 321 | 321
Micrograms*hours per milliliter | 3756.03 [3648.02 to 3867.25] | 2449.75 [2378.56 to 2523.07]

44. Secondary Outcome: AUC for RPV LA
Description: Blood samples were collected at indicated time points to analyze concentration in plasma for RPV LA. Participants who transitioned from ATLAS (201585 - NCT02951052) into this ATLAS-2M (207966) study had been treated with CAB + RPV for at least one year, were approaching steady state exposures, and were therefore excluded in order to focus the population analysis on those without prior exposure.
Time Frame: Predose at Weeks 4, 8, 13, 24, 32, 40, 48; 1 Week post-dose at Week 9 and 41
Population: PK Population. Only those participants with data available at specified time points has been analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Nanograms*hours per milliliter
Arm/Group | RPV LA Q8W | RPV LA Q4W
Number analyzed (Participants) | 321 | 320
Nanograms*hours per milliliter | 126467.59 [122284.26 to 130794.04] | 70306.62 [67814.64 to 72890.17]

45. Secondary Outcome: Maximum Concentration (Cmax) in Plasma for CAB LA Evaluable
Description: Blood samples were collected at indicated time points to analyze Cmax in plasma for CAB LA. Participants who transitioned from ATLAS (201585 - NCT02951052) into this ATLAS-2M (207966) study had been treated with CAB + RPV for at least one year, were approaching steady state exposures, and were therefore excluded in order to focus the population analysis on those without prior exposure.
Time Frame: Predose at Weeks 4, 8, 13, 24, 32, 40, 48; 1 Week post-dose at Week 9 and 41
Population: PK Population. Only those participants with data available at specified time points has been analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Micrograms per milliliter
Arm/Group | CAB LA Q8W | CAB LA Q4W
Number analyzed (Participants) | 321 | 321
Micrograms per milliliter | 3.976 [3.839 to 4.117] | 4.277 [4.140 to 4.418]

46. Secondary Outcome: Cmax in Plasma for RPV LA Evaluable
Description: Blood samples were collected at indicated time points to analyze Cmax in plasma for RPV LA. Participants who transitioned from ATLAS (201585 - NCT02951052) into this ATLAS-2M (207966) study had been treated with CAB + RPV for at least one year, were approaching steady state exposures, and were therefore excluded in order to focus the population analysis on those without prior exposure.
Time Frame: Predose at Weeks 4, 8, 13, 24, 32, 40, 48; 1 Week post-dose at Week 9 and 41
Population: PK Population. Only those participants with data available at specified time points has been analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Nanograms per milliliter
Arm/Group | RPV LA Q8W | RPV LA Q4W
Number analyzed (Participants) | 321 | 320
Nanograms per milliliter | 133.062 [128.452 to 137.837] | 124.279 [119.825 to 128.899]

47. Other Pre Specified Outcome: Number of Participants With Different Demographic Parameters for Inter-participant Variability
Description: Blood samples were planned to be collected at indicated time points for PK analysis of CAB LA and RPV LA. Demographic parameters including, but not limited to, age, sex, race, body weight, body mass index, and relevant laboratory parameters were planned to be evaluated as potential predictors of inter participant variability for pharmacokinetic parameters.
Time Frame: Up to Week 48
Population: PK Population. This was an exploratory Outcome Measure. Data will not be analyzed and reported.
Groups:
- CAB LA: Participants in this arm received CAB LA 600 mg Q8W and 400 mg Q4W through Week 48
- RPV LA: Participants in this arm received RPV LA 900 mg Q8W and 600 mg Q4W through Week 48
Arm/Group | CAB LA | RPV LA
Number analyzed (Participants) | 0 | 0

48. Other Pre Specified Outcome: Number of Participants With Different Demographic Parameters for Intra-participant Variability
Description: Blood samples were planned to be collected at indicated time points for PK analysis of CAB LA and RPV LA. Demographic parameters including, but not limited to, age, sex, race, body weight, body mass index, and relevant laboratory parameters were planned to be evaluated as potential predictors of intra participant variability for pharmacokinetic parameters.
Time Frame: Up to Week 48
Population: PK Population. This was an exploratory Outcome Measure. Data will not be analyzed and reported.
Arm/Group | CAB LA | RPV LA
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Non-SAEs and SAEs were collected from the start of the treatment and up to Week 48 analysis
Description: Non-SAEs and SAEs were collected in Safety Population.
Arm/Group | CAB LA + RPV LA Q8W | CAB LA + RPV LA Q4W
All-Cause Mortality (participants affected / at risk) | 1/522 | 0/523
Serious Adverse Events (participants affected / at risk) | 27/522 | 19/523
Other Adverse Events (participants affected / at risk) | 429/522 | 427/523
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAB LA + RPV LA Q8W (N=522) | CAB LA + RPV LA Q4W (N=523)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2)
Acute hepatitis B (Infections and infestations) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 2 (2) | 0 (0)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0)
Acute hepatitis C (Infections and infestations) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Epiglottitis obstructive (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Gastritis viral (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis Escherichia coli (Infections and infestations) | 1 (1) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0)
Injection site abscess (Infections and infestations) | 1 (1) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Sialoadenitis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oroantral fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic pseudocyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Drug dependence (Psychiatric disorders) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0)
Substance-induced psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Priapism (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAB LA + RPV LA Q8W (N=522) | CAB LA + RPV LA Q4W (N=523)
Injection site pain (General disorders) | 371 (2014) | 363 (2568)
Injection site nodule (General disorders) | 54 (113) | 89 (204)
Injection site induration (General disorders) | 41 (86) | 39 (96)
Injection site discomfort (General disorders) | 36 (92) | 41 (110)
Pyrexia (General disorders) | 28 (46) | 44 (70)
Injection site swelling (General disorders) | 32 (70) | 27 (45)
Injection site pruritus (General disorders) | 27 (63) | 25 (55)
Fatigue (General disorders) | 13 (18) | 33 (41)
Nasopharyngitis (Infections and infestations) | 71 (86) | 74 (101)
Upper respiratory tract infection (Infections and infestations) | 50 (65) | 71 (99)
Gastroenteritis (Infections and infestations) | 16 (17) | 28 (28)
Pharyngitis (Infections and infestations) | 16 (16) | 28 (31)
Headache (Nervous system disorders) | 35 (45) | 36 (53)
Diarrhoea (Gastrointestinal disorders) | 33 (35) | 37 (39)
Back pain (Musculoskeletal and connective tissue disorders) | 28 (32) | 29 (39)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (17) | 29 (30)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-07-03): https://cdn.clinicaltrials.gov/large-docs/49/NCT03299049/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-17): https://cdn.clinicaltrials.gov/large-docs/49/NCT03299049/SAP_001.pdf